CLINICAL TRIAL: NCT02504671
Title: A Phase IIb, Double-Blind, Placebo-Controlled, Dose-Adaptive, Study of the Efficacy and Safety of GSK3196165 in Combination With Methotrexate Therapy, in Subjects With Active Moderate-Severe Rheumatoid Arthritis Despite Treatment With Methotrexate
Brief Title: Study to Evaluate the Efficacy and Safety of GSK3196165 Plus Methotrexate in Subjects With Active Moderate-Severe Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201755; 2014-003453-34 (EudraCT Number)
Record Dates: First submitted 2015-07-20; First posted 2015-07-22 (Estimated); Results first posted 2019-04-04 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2020-12

CONDITIONS: Arthritis, Rheumatoid
Keywords: DMARD-IR; GSK3196165; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Otilimab; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- GSK3196165, Dose 1 + MTX and Folic acid (Experimental): Subject will receive GSK3196165 Dose 1 (initially weekly, then every other week) in combination with MTX (at a dose between 15-25 mg/week) and folic acid >=5 mg/week.
  Interventions: Drug: GSK3196165; Drug: MTX; Drug: Folic acid
- GSK3196165, Dose 2 + MTX and folic acid (Experimental): Subject will receive GSK3196165 Dose 2 (initially weekly, then every other week) in combination with MTX (at a dose between 15-25 mg/week) and folic acid >=5 mg/week.
  Interventions: Drug: GSK3196165; Drug: MTX; Drug: Folic acid
- GSK3196165, Dose 3 + MTX and folic acid (Experimental): Subject will receive GSK3196165 Dose 3 (initially weekly, then every other week) in combination with MTX (at a dose between 15-25 mg/week) and folic acid >=5 mg/week.
  Interventions: Drug: GSK3196165; Drug: MTX; Drug: Folic acid
- GSK3196165, Dose 4 + MTX and folic acid (Experimental): Subject will receive GSK3196165 Dose 4 (initially weekly, then every other week) in combination with MTX (at a dose between 15-25 mg/week) and folic acid >=5 mg/week.
  Interventions: Drug: GSK3196165; Drug: MTX; Drug: Folic acid
- GSK3196165, Dose 5 + MTX and folic acid (Experimental): Subject will receive GSK3196165 Dose 5 (initially weekly, then every other week) in combination with MTX (at a dose between 15-25 mg/week) and folic acid >=5 mg/week.
  Interventions: Drug: GSK3196165; Drug: MTX; Drug: Folic acid
- Placebo + MTX and folic acid (Placebo Comparator): Subjects will receive placebo (initially weekly, then every other week) in combination with MTX (at a dose between 15-25 mg/week) and folic acid >=5 mg/week.
  Interventions: Drug: MTX; Drug: Folic acid; Drug: Placebo

INTERVENTIONS:
Drug: GSK3196165 — GSK3196165 is supplied as liquid and will be administered as SC injection.
  Arms: GSK3196165, Dose 1 + MTX and Folic acid; GSK3196165, Dose 2 + MTX and folic acid; GSK3196165, Dose 3 + MTX and folic acid; GSK3196165, Dose 4 + MTX and folic acid; GSK3196165, Dose 5 + MTX and folic acid
Drug: MTX — MTX will be supplied as capsule, tablet or liquid and will be administered orally or as SC injection.
Drug: Folic acid — Folic acid will be supplied as capsule, tablet or liquid and will be administered orally.
Drug: Placebo — Placebo is supplied as liquid as sterile 0.9% weight by volume (w/v) sodium chloride solution and will be administered as SC injection
  Arms: Placebo + MTX and folic acid

SUMMARY:
This is a randomised, Phase IIb, dose-adaptive, multicentre, double-blind, parallel group, placebo-controlled study with the primary objective to assess the efficacy of GSK3196165, in combination with methotrexate (MTX), in subjects with active moderate severe rheumatoid arthritis (RA) despite treatment with MTX. Approximately 210 subjects will be randomised into the study, following a screening period of up to four weeks. The total treatment period is up to 52 weeks, with a 12-week follow-up period after the last dose (Week 50). Subjects will be randomised (1:1:1:1:1:1) to placebo or one of five subcutaneous (SC) GSK3196165 doses, in combination with MTX (at a weekly dose between 15-25 milligram [mg]), previously received for at least 12 weeks, with a stable and tolerated dose and route of administration for >=4 weeks. Escape therapy is provided at specified timepoints in the protocol for subjects that do not achieve adequate disease improvement.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years at the time of signing informed consent.
* Meets ACR/EULAR 2010 RA Classification Criteria, with disease duration of >=12 weeks.
* Swollen joint count of >=4 (66-joint count) and tender joint count of >=4 (68-joint count).
* DAS28(CRP) >=3.2.
* CRP >=5.0 milligram per litre (mg/L) at screening.
* Must have previously received MTX (15-25 mg weekly) for at least 12 weeks before screening, with no change in route of administration, with a stable and tolerated dose for >=4 weeks prior to Day 1. A stable dose of MTX >=7.5 mg/week is acceptable, if the MTX dose has been reduced for reasons of documented intolerance to MTX, e.g. hepatic or hematologic toxicity, or per local requirement.
* Weight >=45 kilogram (kg).
* Male or female subjects are eligible to participate so long as they meet and agree to abide by the contraceptive criteria.
* Diffusing capacity of the lung for carbon monoxide (DLCO) >=60% predicted; forced expiratory volume in 1 second (FEV1) >=70% predicted
* No evidence of active or latent infection with Mycobacterium tuberculosis (TB).

Exclusion Criteria:

* Pregnant or lactating women.
* History of other inflammatory rheumatological or autoimmune disorders, other than Sjögren's syndrome secondary to RA.
* History of any respiratory disease which (in the opinion of the investigator) would compromise subject safety or the ability of the subject to complete the study (e.g. significant interstitial lung disease, such as pulmonary fibrosis, chronic obstructive pulmonary disease (COPD), moderate-severe asthma, bronchiectasis, previous pulmonary alveolar proteinosis [PAP]).
* Clinically-significant or unstable (in the opinion of the investigator) persistent cough or dyspnea that is unexplained.
* Significant unstable or uncontrolled acute or chronic disease which, in the opinion of the investigator, could confound the results of the study or put the subject at undue risk.
* A history of malignancy.
* Hereditary or acquired immunodeficiency disorder, including immunoglobulin deficiency.
* Current/previous Hepatitis B virus (HBV), Hepatitis C virus (HCV) or human immunodeficiency virus (HIV) 1 or 2 infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2015-07-23 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (55):
- Bulgaria (2):
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Sofia
- Canada (2):
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Barrie
- Czechia (4):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Bruntál
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Uherské Hradiště
- GSK Investigational Site, Tallinn, Estonia
- Germany (4):
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Bad Doberan
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Hungary (3):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Kistarcsa
  - GSK Investigational Site, Veszprém
- Italy (3):
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Bologna
  - GSK Investigational Site, Napoli
- Mexico (4):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Cuernavaca, Morelos
  - GSK Investigational Site, Mérida, Yucatán
  - GSK Investigational Site, San Luis Potosí City
- Poland (8):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Bytom
  - GSK Investigational Site, Grodzisk Mazowiecki
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Torun
  - GSK Investigational Site, Warsaw
- Russia (8):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Omsk
  - GSK Investigational Site, Ryazan
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Tver'
  - GSK Investigational Site, Vladimir
  - GSK Investigational Site, Yaroslavl
- South Africa (3):
  - GSK Investigational Site, Pretoria, Gauteng
  - GSK Investigational Site, Panorama / Cape Town
  - GSK Investigational Site, Stellenbosch
- Spain (2):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Madrid
- Ukraine (9):
  - GSK Investigational Site, Ivano-Frankivsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kryvyi Rih
  - GSK Investigational Site, Lviv
  - GSK Investigational Site, Odesa
  - GSK Investigational Site, Poltava
  - GSK Investigational Site, Sumy
  - GSK Investigational Site, Vinnytsia
  - GSK Investigational Site, Zhytomyr
- United Kingdom (2):
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Leeds

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=20744

REFERENCES:
- [Background] Buckley CD, Simon-Campos JA, Zhdan V, Becker B, Davy K, Fisheleva E, Gupta A, Hawkes C, Inman D, Layton M, Mitchell N, Patel J, Saurigny D, Williamson R, Tak PP. Efficacy, patient-reported outcomes, and safety of the anti-granulocyte macrophage colony-stimulating factor antibody otilimab (GSK3196165) in patients with rheumatoid arthritis: a randomised, phase 2b, dose-ranging study. Lancet Rheumatol. 2020 Nov;2(11):e677-e688. doi: 10.1016/S2665-9913(20)30229-0. Epub 2020 Oct 7. PMID 38279364

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a total of 60 sites in 12 countries: Ukraine (11), Poland (10), Russian Federation (10), Mexico (6), Czech Republic (5), Bulgaria (4), South Africa (3), Hungary (3), Estonia (2), Canada (2), United Kingdom (2), and Germany (2) from 23-July-2015 until 29-December-2017.
Pre-assignment Details: A total of 526 participants were screened of which 304 were screen failures and 222 participants were enrolled in the study.
Groups:
- Placebo: Participants received placebo liquid (sterile 0.9% weight/volume) sodium chloride solution) 0.6 milliliter (mL) drawn into a small (1 mL syringe) administered subcutaneously in the thigh/abdomen up to 52 weeks in combination with methotrexate (MTX) tablets (orally)/liquid (subcutaneous injection) at a dose of 7.5 to 25 milligram (mg)/week and folic acid tablet/capsule (orally) at a dose of >=5 mg/week. MTX was taken as a single weekly dose/ divided weekly dose, folic acid was taken the day after and at least 12 hours following MTX administration. Safety was monitored for 1 hour after the injection, for the first 3 injections, then for 30 minutes thereafter.
- GSK3196165 22.5 mg: Participants received GSK3196165 22.5 mg (0.15 mL) liquid drawn into a small (03 mL/0.5 mL syringe) administered subcutaneously in the thigh/abdomen up to 52 weeks in combination with MTX tablets (orally)/liquid (subcutaneous injection) at a dose of 7.5 to 25 mg/week and folic acid tablet/capsule (orally) at a dose of >=5 mg/week. MTX was taken as a single weekly dose/divided weekly dose, folic acid was taken the day after and at least 12 hours following MTX administration. Safety was monitored for 1 hour after the injection, for the first 3 injections, then for 30 minutes thereafter.
- GSK3196165 45 mg: Participants received GSK3196165 45 mg (0.3 mL) liquid drawn into a small (03 mL/0.5 mL syringe) administered subcutaneously in the thigh/abdomen up to 52 weeks in combination with MTX tablets (orally)/liquid (subcutaneous injection) at a dose of 7.5 to 25 mg/week and folic acid tablet/capsule (orally) at a dose of >=5 mg/week. MTX was taken as a single weekly dose/ divided weekly dose, folic acid was taken the day after and at least 12 hours following MTX administration. Safety was monitored for 1 hour after the injection, for the first 3 injections, then for 30 minutes thereafter.
- GSK3196165 90 mg: Participants received GSK3196165 90 mg (0.6 mL) liquid drawn into a small (1 mL syringe) administered subcutaneously in the thigh/abdomen up to 52 weeks in combination with MTX tablets (orally)/liquid (subcutaneous injection) at a dose of 7.5 to 25 mg/week and folic acid tablet/capsule (orally) at a dose of >=5 mg/week. MTX was taken as a single weekly dose/ divided weekly dose, folic acid was taken the day after and at least 12 hours following MTX administration. Safety was monitored for 1 hour after the injection, for the first 3 injections, then for 30 minutes thereafter.
- GSK3196165 135 mg: Participants received GSK3196165 135 mg (0.9 mL) liquid drawn into a small (1 mL syringe) administered subcutaneously in the thigh/abdomen up to 52 weeks in combination with MTX tablets (orally)/liquid (subcutaneous injection) at a dose of 7.5 to 25 mg/week and folic acid tablet/capsule (orally) at a dose of >=5 mg/week. MTX was taken as a single weekly dose/ divided weekly dose, folic acid was taken the day after and at least 12 hours following MTX administration. Safety was monitored for 1 hour after the injection, for the first 3 injections, then for 30 minutes thereafter.
- GSK3196165 180 mg: Participants received GSK3196165 180 mg (1.2 mL) liquid drawn into a small (2 mL/3 mL syringe) administered subcutaneously in the thigh/abdomen up to 52 weeks in combination with MTX tablets (orally)/liquid (subcutaneous injection) at a dose of 7.5 to 25 mg/week and folic acid tablet/capsule (orally) at a dose of >=5 mg/week. MTX was taken as a single weekly dose/divided weekly dose, folic acid was taken the day after and at least 12 hours following MTX administration. Safety was monitored for 1 hour after the injection, for the first 3 injections, then for 30 minutes thereafter.
Period: Overall Study
Arm/Group | Placebo | GSK3196165 22.5 mg | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 135 mg | GSK3196165 180 mg
Started | 37 | 37 | 37 | 37 | 37 | 37
Completed | 25 | 23 | 27 | 27 | 25 | 23
Not Completed | 12 | 14 | 10 | 10 | 12 | 14
Not completed — Withdrawal by Subject | 1 | 5 | 4 | 4 | 5 | 3
Not completed — Lack of Efficacy | 1 | 3 | 1 | 0 | 4 | 4
Not completed — Adverse Event | 1 | 1 | 0 | 1 | 0 | 2
Not completed — Protocol Violation | 2 | 1 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0 | 0 | 1
Not completed — Protocol defined stopping criteria | 7 | 4 | 3 | 5 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received placebo liquid (sterile 0.9% weight/volume) sodium chloride solution) 0.6 mL drawn into a small (1 mL syringe) administered subcutaneously in the thigh/abdomen up to 52 weeks in combination with MTX tablets (orally)/liquid (subcutaneous injection) at a dose of 7.5 to 25 mg/week and folic acid tablet/capsule (orally) at a dose of >=5 mg/week. MTX was taken as a single weekly dose/divided weekly dose, folic acid was taken the day after and at least 12 hours following MTX administration. Safety was monitored for 1 hour after the injection, for the first 3 injections, then for 30 minutes thereafter.
- GSK3196165 45 mg: Participants received GSK3196165 45 mg (0.3 mL) liquid drawn into a small (03 mL/0.5 mL syringe) administered subcutaneously in the thigh/abdomen up to 52 weeks in combination with MTX tablets (orally)/liquid (subcutaneous injection) at a dose of 7.5 to 25 mg/week and folic acid tablet/capsule (orally) at a dose of >=5 mg/week. MTX was taken as a single weekly dose/divided weekly dose, folic acid was taken the day after and at least 12 hours following MTX administration. Safety was monitored for 1 hour after the injection, for the first 3 injections, then for 30 minutes thereafter.
- GSK3196165 90 mg: Participants received GSK3196165 90 mg (0.6 mL) liquid drawn into a small (1 mL syringe) administered subcutaneously in the thigh/abdomen up to 52 weeks in combination with MTX tablets (orally)/liquid (subcutaneous injection) at a dose of 7.5 to 25 mg/week and folic acid tablet/capsule (orally) at a dose of >=5 mg/week. MTX was taken as a single weekly dose/divided weekly dose, folic acid was taken the day after and at least 12 hours following MTX administration. Safety was monitored for 1 hour after the injection, for the first 3 injections, then for 30 minutes thereafter.
- GSK3196165 135 mg: Participants received GSK3196165 135 mg (0.9 mL) liquid drawn into a small (1 mL syringe) administered subcutaneously in the thigh/abdomen up to 52 weeks in combination with MTX tablets (orally)/liquid (subcutaneous injection) at a dose of 7.5 to 25 mg/week and folic acid tablet/capsule (orally) at a dose of >=5 mg/week. MTX was taken as a single weekly dose/divided weekly dose, folic acid was taken the day after and at least 12 hours following MTX administration. Safety was monitored for 1 hour after the injection, for the first 3 injections, then for 30 minutes thereafter.
- GSK3196165 180 mg: Participants received GSK3196165 180 mg (1.2 mL) liquid drawn into a small (2 mL/3 mL syringe) administered subcutaneous in the thigh/abdomen up to 52 weeks in combination with MTX tablets (orally)/liquid (subcutaneous injection) at a dose of 7.5 to 25 mg/week and folic acid tablet/capsule (orally) at a dose of >=5 mg/week. MTX was taken as a single weekly dose/divided weekly dose, folic acid was taken the day after and at least 12 hours following MTX administration. Safety was monitored for 1 hour after the injection, for the first 3 injections, then for 30 minutes thereafter.
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK3196165 22.5 mg | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 135 mg | GSK3196165 180 mg | Total
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37 | 37 | 222
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.0 (11.33) | 48.4 (11.31) | 52.8 (12.22) | 52.7 (11.28) | 47.1 (10.04) | 52.3 (10.76) | 50.5 (11.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 30 | 33 | 27 | 33 | 29 | 180
  Male | 9 | 7 | 4 | 10 | 4 | 8 | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 2 | 3 | 1 | 2 | 2 | 1 | 11
  Black or African American | 0 | 3 | 0 | 0 | 0 | 0 | 3
  White | 34 | 30 | 35 | 35 | 34 | 35 | 203
  American Indian/ Alaskan Native+White | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Black or African American+White | 0 | 1 | 0 | 0 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Disease Activity Score for 28 Different Joints With C-reactive Protein Value (DAS28{CRP}) Remission (DAS28 <2.6) at Week 24
Description: DAS28 is a modification of the original DAS and is based on a count of 28 swollen and tender joints and is used to evaluate a participant's response to treatment. DAS 28 CRP utilizing joint scores from the following 28 joints: elbows, shoulders, elbow, wrists, metacarpal- phalangeal I-V, proximal interphalangeal I-V and knees and is calculated using the following formula: DAS28 (CRP) = 0.56*√(TJC28) +0.28*√(SJC28)+0.014*GH+0.36*ln(CRP+1)+0.96. Where TJC - Tender joint Count, SJC= Swollen Joint Count, (GH=participant assessment of disease activity using a 100 millimeter [mm] visual analogue scale with 0 = best, 100 = worst) and CRP= C reactive Protein (in [milligrams/liter] mg/L). It ranges between 0.96 and 8.61. High score (worse outcome) and low scores (better outcome). ITT population comprised of all participants who were randomized to treatment and who received at least one dose of study treatment (GSK3196165 or placebo).
Time Frame: Week 24
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GSK3196165 22.5 mg | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 135 mg | GSK3196165 180 mg
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37 | 37
Percentage of participants | 3 | 5 | 16 | 19 | 14 | 14
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.547, Regression, Logistic; Odds Ratio (OR) = 2.12, 95% CI 2-sided [0.18 to 24.52] — 95% Confidence Intervals (CI) were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.077, Regression, Logistic; Odds Ratio (OR) = 7.11, 95% CI 2-sided [0.81 to 62.44] — 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.053, Regression, Logistic; Odds Ratio (OR) = 8.39, 95% CI 2-sided [0.98 to 72.14] — 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.122, Regression, Logistic; Odds Ratio (OR) = 5.69, 95% CI 2-sided [0.63 to 51.40] — 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 5: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.134, Regression, Logistic; Odds Ratio (OR) = 5.40, 95% CI 2-sided [0.60 to 48.83] — 95% CI were constructed using asymptotic Wald confidence limits without correction

2. Secondary Outcome: Change From Baseline in DAS28(CRP) at Week 12
Description: DAS28 is a modification of the original DAS and is based on a count of 28 swollen and tender joints and is used to evaluate a participant's response to treatment. DAS 28 CRP utilizing joint scores from the following 28 joints: elbows, shoulders, elbow, wrists, metacarpal- phalangeal I-V, proximal interphalangeal I-V and knees and is calculated using the following formula: DAS28 (CRP) = 0.56*√(TJC28) +0.28*√(SJC28)+0.014*GH+0.36*ln(CRP+1)+0.96. Where TJC - Tender joint Count, SJC= Swollen Joint Count, (GH=participant global assessment of disease activity (PtGA) using a 100 mm visual analogue scale with 0 = best, 100 = worst) and CRP= C reactive Protein (in mg/L). It ranges between 0.96 and 8.61. High score (worse outcome) and low scores (better outcome). Baseline was defined as the last available assessment prior to the start of study treatment. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline and Week 12
Population: ITT Population. Only those participants with data available at the indicated time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | GSK3196165 22.5 mg | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 135 mg | GSK3196165 180 mg
Number analyzed (Participants) | 34 | 35 | 33 | 37 | 34 | 36
Scores on a scale
  CRP | -5.21 (2.730) | -4.75 (2.701) | -8.57 (2.749) | -7.79 (2.624) | -7.71 (2.722) | -7.21 (2.659)
  PtGA | -6.72 (3.660) | -14.40 (3.653) | -20.40 (3.611) | -24.11 (3.544) | -19.35 (3.614) | -23.90 (3.606)
  SJC28 | -2.35 (1.093) | -4.77 (1.085) | -5.52 (1.080) | -6.91 (1.056) | -5.33 (1.080) | -8.39 (1.070)
  TJC28 | -2.81 (1.191) | -5.11 (1.181) | -6.73 (1.173) | -8.53 (1.151) | -6.43 (1.175) | -9.13 (1.167)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.905, Mixed Model Repeated Measures (MMRM) — MMRM analysis adjusted for DAS28(CRP) Baseline score, treatment group, visit and treatment group by visit and Baseline by visit interactions; Mean Difference (Net) = 0.46, 95% CI 2-sided [-7.13 to 8.05] — CRP, Week 12
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.387, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -3.36, 95% CI 2-sided [-11.00 to 4.28] — CRP, Week 12
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.495, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -2.58, 95% CI 2-sided [-10.04 to 4.87] — CRP, Week 12
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.140, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -7.68, 95% CI 2-sided [-17.92 to 2.55] — PtGA, Week 12
Statistical Analysis 5: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.009, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -13.68, 95% CI 2-sided [-23.85 to -3.52] — PtGA, Week 12
Statistical Analysis 6: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -17.40, 95% CI 2-sided [-27.44 to -7.35] — PtGA, Week 12
Statistical Analysis 7: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.118, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -2.42, 95% CI 2-sided [-5.45 to 0.62] — SJC28, Week 12
Statistical Analysis 8: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.041, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -3.17, 95% CI 2-sided [-6.20 to -0.14] — SJC28, Week 12
Statistical Analysis 9: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.003, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -4.56, 95% CI 2-sided [-6.00 to 0.05] — SJC28, Week 12
Statistical Analysis 10: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.172, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -2.30, 95% CI 2-sided [-5.61 to 1.01] — TC28, Week 12
Statistical Analysis 11: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.020, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -3.92, 95% CI 2-sided [-7.22 to -0.62] — TJC28, Week 12
Statistical Analysis 12: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -5.72, 95% CI 2-sided [-8.98 to -2.45] — TJC28, Week 12
Statistical Analysis 13: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.518, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -2.51, 95% CI 2-sided [-10.13 to 5.12] — CRP, Week 12
Statistical Analysis 14: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.599, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -2.00, 95% CI 2-sided [-9.50 to 5.49] — CRP, Week 12
Statistical Analysis 15: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.015, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -12.63, 95% CI 2-sided [-22.78 to -2.48] — PtGA, Week 12
Statistical Analysis 16: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -17.18, 95% CI 2-sided [-27.27 to -7.10] — PtGA, Week 12
Statistical Analysis 17: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.054, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -2.98, 95% CI 2-sided [-6.00 to 0.05] — SJC28, Week 12
Statistical Analysis 18: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -6.04, 95% CI 2-sided [-9.05 to -3.02] — SJC28, Week 12
Statistical Analysis 19: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.031, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -3.63, 95% CI 2-sided [-6.92 to -0.33] — TJC28, Week 12
Statistical Analysis 20: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -6.32, 95% CI 2-sided [-9.61 to -3.02] — TJC28, Week 12

3. Secondary Outcome: Percentage of Participants Who Achieved DAS28(CRP) Remission (DAS28 <2.6) at All Time Points
Description: DAS28(CRP) remission is defined as a DAS28 score of <2.6 points. The DAS index combines information relating to the number of swollen and tender joints. The DAS28 is a modification of the original DAS and is based on a count of 28 swollen and tender joints and is used to evaluate a participant's response to treatment. DAS 28 CRP utilizing joint scores from the following 28 joints: elbows, shoulders, elbow, wrists, metacarpal- phalangeal I-V, proximal interphalangeal I-V and knees and is calculated using the following formula: DAS28 (CRP) = 0.56*√(TJC28) +0.28*√(SJC28)+0.014*GH+0.36*ln(CRP+1)+0.96. Where TJC - Tender joint Count, SJC= Swollen Joint Count, (GH=participant assessment of disease activity using a 100 mm visual analogue scale with 0 = best, 100 = worst) and CRP= C reactive Protein (in mg/L). It ranges between 0.96 and 8.61. High score (worse outcome) and low scores (better outcome).
Time Frame: Weeks 1, 2, 4, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and Week 62 (follow-up)
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GSK3196165 22.5 mg | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 135 mg | GSK3196165 180 mg
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37 | 37
Percentage of participants
  Week 1 | 0 | 0 | 0 | 0 | 0 | 0
  Week 2 | 0 | 0 | 0 | 0 | 0 | 1
  Week 4 | 0 | 0 | 0 | 5 | 3 | 4
  Week 6 | 5 | 5 | 0 | 5 | 3 | 8
  Week 8 | 3 | 0 | 5 | 14 | 5 | 8
  Week 12 | 3 | 8 | 5 | 24 | 3 | 16
  Week 16 | 0 | 3 | 14 | 27 | 5 | 19
  Week 20 | 3 | 0 | 16 | 19 | 14 | 16
  Week 24 | 3 | 5 | 16 | 19 | 14 | 14
  Week 28 | 3 | 3 | 16 | 16 | 14 | 22
  Week 32 | 3 | 5 | 22 | 14 | 11 | 19
  Week 36 | 3 | 5 | 19 | 8 | 16 | 19
  Week 40 | 0 | 5 | 14 | 14 | 11 | 24
  Week 44 | 3 | 5 | 14 | 16 | 14 | 16
  Week 48 | 0 | 5 | 14 | 14 | 14 | 19
  Week 52 | 3 | 5 | 14 | 11 | 14 | 14
  Week 62 (follow-up) | 3 | 0 | 8 | 3 | 11 | 19
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — Week 4. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 0.0, 95% CI 2-sided [-10.3 to 10.3] — Week 6. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = -5.4, 95% CI 2-sided [-12.7 to 1.9] — Week 6. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 0.0, 95% CI 2-sided [-10.3 to 10.3] — Week 6. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 5: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = -2.7, 95% CI 2-sided [-7.9 to 2.5] — Week 8. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 6: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-6.3 to 11.7] — Week 8. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 7: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [-1.4 to 23.0] — Week 8. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 8: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-4.8 to 15.6] — Week 12. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 9: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-6.3 to 11.7] — Week 12. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 10: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 21.6, 95% CI 2-sided [6.8 to 36.4] — Week 12. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 11: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — Week 16. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 12: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [2.5 to 24.5] — Week 16. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 13: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 27.0, 95% CI 2-sided [12.7 to 41.3] — Week 16. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 14: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = -2.7, 95% CI 2-sided [-7.9 to 2.5] — Week 20. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 15: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — Week 20. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 16: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [2.6 to 29.9] — Week 20. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 17: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-6.3 to 11.7] — Week 24. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 18: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — Week 24. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 19: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [2.6 to 29.9] — Week 24. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 20: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 0.0, 95% CI 2-sided [-7.4 to 7.4] — Week 28. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 21: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — Week 28. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 22: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — Week 28. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 23: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-6.3 to 11.7] — Week 32. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 24: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 18.9, 95% CI 2-sided [4.7 to 33.2] — Week 32. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 25: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [-1.4 to 23.0] — Week 32. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 26: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-6.3 to 11.7] — Week 36. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 27: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [2.6 to 29.9] — Week 36. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 28: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-4.8 to 15.6] — Week 36. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 29: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — Week 40. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 30: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [2.5 to 24.5] — Week 40. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 31: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [2.5 to 24.5] — Week 40. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 32: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-6.3 to 11.7] — Week 44. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 33: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [-1.4 to 23.0] — Week 44. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 34: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — Week 44. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 35: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — Week 48. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 36: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [2.5 to 24.5] — Week 48. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 37: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [2.5 to 24.5] — Week 48. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 38: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-6.3 to 11.7] — Week 52. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 39: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [-1.4 to 23.0] — Week 52. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 40: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-3.2 to 19.4] — Week 52. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 41: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = -2.7, 95% CI 2-sided [-7.9 to 2.5] — Week 62 (follow-up). 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 42: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-4.8 to 15.6] — Week 62 (follow-up). 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 43: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 0.0, 95% CI 2-sided [-7.4 to 7.4] — Week 62 (follow-up). 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 44: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — Week 2. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 45: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — Week 4. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 46: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [0.8 to 20.8] — Week 4. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 47: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = -2.7, 95% CI 2-sided [-11.7 to 6.3] — 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 48: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-8.7 to 14.1] — Week 6. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 49: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-6.3 to 11.7] — Week 8. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 50: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-4.8 to 15.6] — Week 8. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 51: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 0.0, 95% CI 2-sided [-7.4 to 7.4] — Week 12. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 52: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — Week 12. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 53: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — Week 16. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 54: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 18.9, 95% CI 2-sided [6.3 to 31.5] — Week 16. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 55: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [-1.4 to 23.0] — Week 20. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 56: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — Week 20. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 57: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [-1.4 to 23.0] — Week 24. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 58: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [-1.4 to 23.0] — Week 24. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 59: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [-1.4 to 23.0] — Week 28. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 60: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 18.9, 95% CI 2-sided [4.7 to 33.2] — Week 28. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 61: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-3.2 to 19.4] — Week 32. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 62: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [2.6 to 29.9] — Week 32. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 63: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — Week 36. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 64: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [2.6 to 29.9] — Week 36, 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 65: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [0.8 to 20.8] — Week 40. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 66: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 24.3, 95% CI 2-sided [10.5 to 38.1] — Week 40. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 67: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [-1.4 to 23.0] — Week 44. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 68: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — Week 44. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 69: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [2.5 to 24.5] — Week 48. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 70: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 18.9, 95% CI 2-sided [6.3 to 31.5] — Week 48. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 71: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [-1.4 to 23.0] — Week 52. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 72: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [-1.4 to 23.0] — Week 52. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 73: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-3.2 to 19.4] — Week 62 (follow-up). 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 74: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [2.6 to 29.9] — Week 62 (follow-up). 95% CI were constructed using asymptotic Wald confidence limits without correction

4. Secondary Outcome: Change From Baseline in DAS28(CRP) at All Assessment Time Points
Description: DAS28 is a modification of the original DAS and is based on a count of 28 swollen and tender joints and is used to evaluate a participant's response to treatment. DAS 28 CRP utilizing joint scores from the following 28 joints: elbows, shoulders, elbow, wrists, metacarpal- phalangeal I-V, proximal interphalangeal I-V and knees and is calculated using the following formula: DAS28 (CRP) = 0.56*√(TJC28) +0.28*√(SJC28)+0.014*GH+0.36*ln(CRP+1)+0.96. Where TJC - Tender joint Count, SJC= Swollen Joint Count, (GH=participant assessment of disease activity using a 100 mm visual analogue scale with 0 = best, 100 = worst) and CRP= C reactive Protein (in mg/L). It ranges between 0.96 and 8.61. High score (worse outcome) and low scores (better outcome). Baseline was defined as the last available assessment prior to the start of study treatment. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline.
Time Frame: Baseline and Weeks 1, 2, 4, 6, 8, 12, 16, 20 and 24
Population: ITT Population. Only those participants with data available at specified time points were analyzed (indicated by n=X in category titles).
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | GSK3196165 22.5 mg | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 135 mg | GSK3196165 180 mg
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37 | 37
Scores on a scale
  Week 1; n=35, 36, 33, 35, 34, 37: number analyzed (Participants) | 35 | 36 | 33 | 35 | 34 | 37
  Week 1; n=35, 36, 33, 35, 34, 37 | -0.14 (0.114) | -0.47 (0.114) | -0.44 (0.117) | -0.52 (0.114) | -0.55 (0.116) | -0.63 (0.112)
  Week 2; n=36, 35, 34, 36, 36, 36: number analyzed (Participants) | 36 | 35 | 34 | 36 | 36 | 36
  Week 2; n=36, 35, 34, 36, 36, 36 | -0.37 (0.138) | -0.64 (0.141) | -0.69 (0.142) | -0.78 (0.138) | -0.84 (0.139) | -0.88 (0.139)
  Week 4; n=32, 33, 34, 36, 36, 36: number analyzed (Participants) | 32 | 33 | 34 | 36 | 36 | 36
  Week 4; n=32, 33, 34, 36, 36, 36 | -0.45 (0.169) | -0.85 (0.169) | -1.01 (0.167) | -1.21 (0.163) | -1.12 (0.164) | -1.46 (0.164)
  Week 6; n=35, 34, 34, 36, 33, 36: number analyzed (Participants) | 35 | 34 | 34 | 36 | 33 | 36
  Week 6; n=35, 34, 34, 36, 33, 36 | -0.65 (0.184) | -1.07 (0.186) | -1.12 (0.185) | -1.26 (0.181) | -1.12 (0.185) | -1.51 (0.182)
  Week 8; n=34, 33, 34, 37, 35, 32: number analyzed (Participants) | 34 | 33 | 34 | 37 | 35 | 32
  Week 8; n=34, 33, 34, 37, 35, 32 | -0.61 (0.195) | -1.04 (0.197) | -1.40 (0.196) | -1.44 (0.190) | -1.51 (0.194) | -1.72 (0.196)
  Week 12; n=34, 35, 33, 37, 34, 36: number analyzed (Participants) | 34 | 35 | 33 | 37 | 34 | 36
  Week 12; n=34, 35, 33, 37, 34, 36 | -0.60 (0.232) | -1.13 (0.231) | -1.48 (0.233) | -1.84 (0.225) | -1.28 (0.230) | -1.87 (0.228)
  Week 16; n=8, 16, 20, 24, 18, 36: number analyzed (Participants) | 8 | 16 | 20 | 24 | 18 | 36
  Week 16; n=8, 16, 20, 24, 18, 36 | -0.87 (0.335) | -1.16 (0.274) | -1.86 (0.261) | -1.88 (0.247) | -1.64 (0.265) | -1.98 (0.232)
  Week 20; n=8, 15, 20, 25, 19, 36: number analyzed (Participants) | 8 | 15 | 20 | 25 | 19 | 36
  Week 20; n=8, 15, 20, 25, 19, 36 | -1.23 (0.359) | -1.30 (0.284) | -1.81 (0.260) | -1.89 (0.241) | -2.00 (0.263) | -2.03 (0.221)
  Week 24; n=8, 14, 20, 24, 19, 33: number analyzed (Participants) | 8 | 14 | 20 | 24 | 19 | 33
  Week 24; n=8, 14, 20, 24, 19, 33 | -0.23 (0.402) | -1.45 (0.322) | -1.76 (0.288) | -1.62 (0.269) | -1.71 (0.291) | -2.05 (0.246)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.046, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.32, 95% CI 2-sided [-0.64 to -0.01] — Week 1
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.071, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.30, 95% CI 2-sided [-0.62 to 0.03] — Week 1
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.022, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.37, 95% CI 2-sided [-0.69 to -0.05] — Week 1
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.160, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.28, 95% CI 2-sided [-0.67 to 0.11] — Week 2
Statistical Analysis 5: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.103, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.32, 95% CI 2-sided [-0.71 to 0.07] — Week 2
Statistical Analysis 6: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.034, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.42, 95% CI 2-sided [-0.80 to -0.03] — Week 2
Statistical Analysis 7: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.096, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.40, 95% CI 2-sided [-0.87 to 0.07] — Week 4
Statistical Analysis 8: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.020, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.56, 95% CI 2-sided [-1.02 to -0.09] — Week 4
Statistical Analysis 9: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.76, 95% CI 2-sided [-1.22 to -0.29] — Week 4
Statistical Analysis 10: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.110, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.42, 95% CI 2-sided [-0.93 to 0.10] — Week 6
Statistical Analysis 11: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.076, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.47, 95% CI 2-sided [-0.98 to 0.05] — Week 6
Statistical Analysis 12: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.020, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.61, 95% CI 2-sided [-1.11 to -0.10] — Week 6
Statistical Analysis 13: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.128, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.42, 95% CI 2-sided [-0.97 to 0.12] — Week 8
Statistical Analysis 14: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.005, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.78, 95% CI 2-sided [-1.33 to -0.24] — Week 8
Statistical Analysis 15: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.003, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.82, 95% CI 2-sided [-1.36 to -0.29] — Week 8
Statistical Analysis 16: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.110, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.53, 95% CI 2-sided [-1.17 to 0.12] — Week 12
Statistical Analysis 17: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.008, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.88, 95% CI 2-sided [-1.53 to -0.23] — Week 12
Statistical Analysis 18: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -1.24, 95% CI 2-sided [-1.88 to -0.60] — Week 12
Statistical Analysis 19: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.500, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.29, 95% CI 2-sided [-1.15 to 0.56] — Week 16
Statistical Analysis 20: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.021, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.99, 95% CI 2-sided [-1.83 to -0.15] — Week 16
Statistical Analysis 21: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.017, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -1.00, 95% CI 2-sided [-1.83 to -0.18] — Week 16
Statistical Analysis 22: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.871, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.98 to 0.83] — Week 20
Statistical Analysis 23: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.190, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.58, 95% CI 2-sided [-1.46 to 0.29] — Week 20
Statistical Analysis 24: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.130, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.66, 95% CI 2-sided [-1.51 to 0.20] — Week 20
Statistical Analysis 25: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.019, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -1.22, 95% CI 2-sided [-2.24 to -0.20] — Week 24
Statistical Analysis 26: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.002, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -1.53, 95% CI 2-sided [-2.51 to -0.55] — Week 24
Statistical Analysis 27: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.005, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -1.39, 95% CI 2-sided [-2.34 to -0.43] — Week 24
Statistical Analysis 28: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.013, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.41, 95% CI 2-sided [-0.73 to -0.09] — Week 1
Statistical Analysis 29: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.003, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.49, 95% CI 2-sided [-0.80 to -0.17] — Week 1
Statistical Analysis 30: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.017, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.47, 95% CI 2-sided [-0.86 to -0.09] — Week 2
Statistical Analysis 31: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.009, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.52, 95% CI 2-sided [-0.90 to -0.13] — Week 2
Statistical Analysis 32: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.005, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.67, 95% CI 2-sided [-1.13 to -0.20] — Week 4
Statistical Analysis 33: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -1.01, 95% CI 2-sided [-1.48 to -0.55] — Week 4
Statistical Analysis 34: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.073, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.47, 95% CI 2-sided [-0.99 to 0.04] — Week 6
Statistical Analysis 35: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.85, 95% CI 2-sided [-1.36 to -0.34] — Week 6
Statistical Analysis 36: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.89, 95% CI 2-sided [-1.43 to -0.35] — Week 8
Statistical Analysis 37: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -1.10, 95% CI 2-sided [-1.65 to -0.56] — Week 8
Statistical Analysis 38: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.039, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.68, 95% CI 2-sided [-1.32 to -0.03] — Week 12
Statistical Analysis 39: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -1.27, 95% CI 2-sided [-1.91 to -0.63] — Week 12
Statistical Analysis 40: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.073, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.77, 95% CI 2-sided [-1.61 to 0.07] — Week 16
Statistical Analysis 41: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.007, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -1.11, 95% CI 2-sided [-1.91 to -0.30] — Week 16
Statistical Analysis 42: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.083, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.77, 95% CI 2-sided [-1.65 to 0.10] — Week 20
Statistical Analysis 43: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.059, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.80, 95% CI 2-sided [-1.63 to 0.03] — Week 20
Statistical Analysis 44: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.003, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -1.48, 95% CI 2-sided [-2.46 to -0.50] — Week 24
Statistical Analysis 45: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -1.82, 95% CI 2-sided [-2.75 to -0.89] — Week 24

5. Secondary Outcome: Time to First DAS28(CRP) Remission
Description: The DAS index combines information relating to the number of swollen and tender joints. The DAS28 is a modification of the original DAS and is based on a count of 28 swollen and tender joints and is used to evaluate a participant's response to treatment. DAS 28 CRP utilizing joint scores from the following 28 joints: elbows, shoulders, elbow, wrists, metacarpal- phalangeal I-V, proximal interphalangeal I-V and knees and is calculated using the following formula: DAS28 (CRP) = 0.56*√(TJC28) +0.28*√(SJC28)+0.014*GH+0.36*ln(CRP+1)+0.96. Where TJC - Tender joint Count, SJC= Swollen Joint Count, (GH=participant assessment of disease activity using a 100 mm visual analogue scale with 0 = best, 100 = worst) and CRP= C reactive Protein (in mg/L). It ranges between 0.96 and 8.61. High score (worse outcome) and low scores (better outcome). Median time, to remission has been presented.
Time Frame: Up to Week 62
Population: ITT Population. Only those participants with data available at the time of assessment were analyzed.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Placebo | GSK3196165 22.5 mg | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 135 mg | GSK3196165 180 mg
Number analyzed (Participants) | 4 | 6 | 11 | 10 | 7 | 18
Weeks | 9.10 [6.0 to 20.3] | 12.05 [6.1 to 24.3] | 16.10 [8.0 to 24.9] | 8.10 [4.1 to 16.3] | 19.90 [4.3 to 24.9] | 18.20 [2.0 to 64.1]

6. Secondary Outcome: Percentage of Participants Achieving Categorical DAS28(CRP) Response (Moderate/Good [European League Against Rheumatism] EULAR Response) at All Assessment Time Points
Description: DAS28(CRP) scores were categorized using EULAR response criteria. Response at a given time point was defined based on the combination of current DAS28 score and the improvement in the current DAS28 score relative to Baseline. The definition of no response, moderate response and good response was as follows: Current DAS28 <=3.2 and DAS28 decrease from Baseline (>1.2=good response), (>0.6 to <=1.2 = moderate response) and (<=0.6 =no response). Current DAS28 >3.2 to <=5.1 and DAS28 decrease from Baseline value (>1.2 =moderate response), (>0.6 to <=1.2 = moderate response) and (<=0.6 =no response). Current DAS28 >5.1 and DAS28 decrease from Baseline value (>1.2=moderate response), (>0.6 to <=1.2 = no response) and (<=0.6 =no response). If the post-Baseline DAS28(CRP) score was missing, then the corresponding EULAR category was set to missing.
Time Frame: Weeks 1, 2, 4, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and Week 62 (follow-up)
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GSK3196165 22.5 mg | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 135 mg | GSK3196165 180 mg
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37 | 37
Percentage of participants
  Week 1 | 5 | 22 | 16 | 24 | 19 | 27
  Week 2 | 14 | 19 | 16 | 38 | 32 | 38
  Week 4 | 16 | 46 | 38 | 46 | 43 | 68
  Week 6 | 24 | 46 | 43 | 51 | 46 | 65
  Week 8 | 32 | 43 | 59 | 65 | 59 | 68
  Week 12 | 22 | 43 | 51 | 68 | 49 | 76
  Week 16 | 22 | 35 | 54 | 59 | 43 | 73
  Week 20 | 16 | 35 | 51 | 65 | 43 | 73
  Week 24 | 16 | 32 | 46 | 54 | 43 | 70
  Week 28 | 3 | 8 | 19 | 19 | 16 | 78
  Week 32 | 3 | 8 | 22 | 22 | 16 | 73
  Week 36 | 3 | 8 | 19 | 22 | 16 | 73
  Week 40 | 3 | 8 | 19 | 22 | 16 | 65
  Week 44 | 3 | 8 | 19 | 19 | 16 | 59
  Week 48 | 3 | 8 | 19 | 19 | 16 | 65
  Week 52 | 3 | 8 | 16 | 16 | 16 | 51
  Week 62 (follow-up) | 3 | 5 | 16 | 16 | 16 | 54
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.037, Regression, Logistic; Difference = 16.2, 95% CI 2-sided [1.1 to 31.4] — Difference to placebo for Week 1 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.144, Regression, Logistic; Difference = 10.8, 95% CI 2-sided [-3.1 to 24.7] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.033, Regression, Logistic; Difference = 18.9, 95% CI 2-sided [3.3 to 34.5] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.437, Regression, Logistic; Difference = 5.4, 95% CI 2-sided [-11.3 to 22.2] — Difference to placebo for Week 2 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 5: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.755, Regression, Logistic; Difference = 2.7, 95% CI 2-sided [-13.5 to 18.9] — [estimate comment as in outcome 6, analysis 4]
Statistical Analysis 6: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.023, Regression, Logistic; Difference = 24.3, 95% CI 2-sided [5.2 to 43.4] — [estimate comment as in outcome 6, analysis 4]
Statistical Analysis 7: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.006, Regression, Logistic; Difference = 29.7, 95% CI 2-sided [9.8 to 49.7] — Difference to placebo for Week 4 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 8: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.039, Regression, Logistic; Difference = 21.6, 95% CI 2-sided [2.0 to 41.2] — [estimate comment as in outcome 6, analysis 7]
Statistical Analysis 9: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.008, Regression, Logistic; Difference = 29.7, 95% CI 2-sided [9.8 to 49.7] — [estimate comment as in outcome 6, analysis 7]
Statistical Analysis 10: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.044, Regression, Logistic; Difference = 21.6, 95% CI 2-sided [0.4 to 42.8] — [estimate comment as in outcome 6, analysis 7]
Statistical Analysis 11: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.083, Regression, Logistic; Difference = 18.9, 95% CI 2-sided [-2.2 to 40.0] — Difference to placebo for Week 6 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 12: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 27.0, 95% CI 2-sided [5.8 to 48.3] — [estimate comment as in outcome 6, analysis 11]
Statistical Analysis 13: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [-11.2 to 32.8] — Difference to placebo for Week 8 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction.Wald confidence limits without correction
Statistical Analysis 14: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 27.0, 95% CI 2-sided [5.2 to 48.9] — Difference to placebo for Week 8 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 15: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 32.4, 95% CI 2-sided [10.9 to 54.0] — [estimate comment as in outcome 6, analysis 14]
Statistical Analysis 16: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 21.6, 95% CI 2-sided [0.9 to 42.4] — Difference to placebo for Week 12 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 17: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 29.7, 95% CI 2-sided [8.9 to 50.6] — [estimate comment as in outcome 6, analysis 16]
Statistical Analysis 18: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 45.9, 95% CI 2-sided [25.9 to 66.0] — [estimate comment as in outcome 6, analysis 16]
Statistical Analysis 19: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [-6.8 to 33.8] — Difference to placebo for Week 16 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 20: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 32.4, 95% CI 2-sided [11.6 to 53.3] — [estimate comment as in outcome 6, analysis 19]
Statistical Analysis 21: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 37.8, 95% CI 2-sided [17.2 to 58.5] — [estimate comment as in outcome 6, analysis 19]
Statistical Analysis 22: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 18.9, 95% CI 2-sided [-0.5 to 38.4] — Difference to placebo for Week 20 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 23: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 35.1, 95% CI 2-sided [15.1 to 55.1] — [estimate comment as in outcome 6, analysis 22]
Statistical Analysis 24: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 48.6, 95% CI 2-sided [29.2 to 68.1] — [estimate comment as in outcome 6, analysis 22]
Statistical Analysis 25: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [-3.0 to 35.4] — Difference to placebo for Week 24 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 26: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 29.7, 95% CI 2-sided [9.8 to 49.7] — [estimate comment as in outcome 6, analysis 25]
Statistical Analysis 27: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 37.8, 95% CI 2-sided [17.9 to 57.8] — [estimate comment as in outcome 6, analysis 25]
Statistical Analysis 28: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-4.8 to 15.6] — Difference to placebo for Week 28 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 29: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [2.6 to 29.9] — [estimate comment as in outcome 6, analysis 28]
Statistical Analysis 30: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [2.6 to 29.9] — [estimate comment as in outcome 6, analysis 28]
Statistical Analysis 31: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-4.8 to 15.6] — Difference to placebo for Week 32 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 32: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 18.9, 95% CI 2-sided [4.7 to 33.2] — [estimate comment as in outcome 6, analysis 31]
Statistical Analysis 33: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 18.9, 95% CI 2-sided [4.7 to 33.2] — [estimate comment as in outcome 6, analysis 31]
Statistical Analysis 34: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-4.8 to 15.6] — Difference to placebo for Week 36 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 35: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [2.6 to 29.9] — [estimate comment as in outcome 6, analysis 34]
Statistical Analysis 36: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 18.9, 95% CI 2-sided [4.7 to 33.2] — [estimate comment as in outcome 6, analysis 34]
Statistical Analysis 37: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-4.8 to 15.6] — Difference to placebo for Week 40 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 38: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [2.6 to 29.9] — [estimate comment as in outcome 6, analysis 37]
Statistical Analysis 39: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 18.9, 95% CI 2-sided [4.7 to 33.2] — [estimate comment as in outcome 6, analysis 37]
Statistical Analysis 40: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-4.8 to 15.6] — Difference to placebo for Week 48 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 41: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [2.6 to 29.9] — [estimate comment as in outcome 6, analysis 40]
Statistical Analysis 42: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [2.6 to 29.9] — [estimate comment as in outcome 6, analysis 40]
Statistical Analysis 43: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-4.8 to 15.6] — Difference to placebo for Week 52 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 44: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — [estimate comment as in outcome 6, analysis 43]
Statistical Analysis 45: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — [estimate comment as in outcome 6, analysis 43]
Statistical Analysis 46: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-6.3 to 11.7] — Difference to placebo for Week 62 (follow-up) is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 47: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — [estimate comment as in outcome 6, analysis 46]
Statistical Analysis 48: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — [estimate comment as in outcome 6, analysis 46]
Statistical Analysis 49: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [-1.1 to 28.1] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 50: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 21.6, 95% CI 2-sided [5.6 to 37.7] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 51: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 18.9, 95% CI 2-sided [0.2 to 37.6] — [estimate comment as in outcome 6, analysis 4]
Statistical Analysis 52: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 24.3, 95% CI 2-sided [5.2 to 43.4] — [estimate comment as in outcome 6, analysis 4]
Statistical Analysis 53: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 27.0, 95% CI 2-sided [7.1 to 46.9] — [estimate comment as in outcome 6, analysis 7]
Statistical Analysis 54: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 51.4, 95% CI 2-sided [32.2 to 70.5] — [estimate comment as in outcome 6, analysis 7]
Statistical Analysis 55: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 21.6, 95% CI 2-sided [0.4 to 42.8] — [estimate comment as in outcome 6, analysis 11]
Statistical Analysis 56: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 40.5, 95% CI 2-sided [19.9 to 61.2] — [estimate comment as in outcome 6, analysis 11]
Statistical Analysis 57: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 27.0, 95% CI 2-sided [5.2 to 48.9] — [estimate comment as in outcome 6, analysis 14]
Statistical Analysis 58: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 35.1, 95% CI 2-sided [13.8 to 56.5] — [estimate comment as in outcome 6, analysis 14]
Statistical Analysis 59: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 27.0, 95% CI 2-sided [6.2 to 47.9] — [estimate comment as in outcome 6, analysis 16]
Statistical Analysis 60: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 54.1, 95% CI 2-sided [34.9 to 73.2] — [estimate comment as in outcome 6, analysis 16]
Statistical Analysis 61: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 21.6, 95% CI 2-sided [0.9 to 42.4] — [estimate comment as in outcome 6, analysis 19]
Statistical Analysis 62: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 51.4, 95% CI 2-sided [31.8 to 70.9] — [estimate comment as in outcome 6, analysis 19]
Statistical Analysis 63: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 27.0, 95% CI 2-sided [7.1 to 46.9] — [estimate comment as in outcome 6, analysis 22]
Statistical Analysis 64: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 56.8, 95% CI 2-sided [38.2 to 75.4] — [estimate comment as in outcome 6, analysis 22]
Statistical Analysis 65: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 27.0, 95% CI 2-sided [7.1 to 46.9] — [estimate comment as in outcome 6, analysis 25]
Statistical Analysis 66: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 54.1, 95% CI 2-sided [35.1 to 73.0] — [estimate comment as in outcome 6, analysis 25]
Statistical Analysis 67: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — [estimate comment as in outcome 6, analysis 28]
Statistical Analysis 68: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 75.7, 95% CI 2-sided [61.4 to 89.9] — [estimate comment as in outcome 6, analysis 28]
Statistical Analysis 69: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — [estimate comment as in outcome 6, analysis 31]
Statistical Analysis 70: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 70.3, 95% CI 2-sided [55.0 to 85.5] — [estimate comment as in outcome 6, analysis 31]
Statistical Analysis 71: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — [estimate comment as in outcome 6, analysis 34]
Statistical Analysis 72: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 70.3, 95% CI 2-sided [55.0 to 85.5] — [estimate comment as in outcome 6, analysis 34]
Statistical Analysis 73: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — [estimate comment as in outcome 6, analysis 37]
Statistical Analysis 74: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 62.2, 95% CI 2-sided [45.9 to 78.4] — [estimate comment as in outcome 6, analysis 37]
Statistical Analysis 75: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — Difference to placebo for Week 44 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 76: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 56.8, 95% CI 2-sided [40.1 to 73.4] — [estimate comment as in outcome 6, analysis 75]
Statistical Analysis 77: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — [estimate comment as in outcome 6, analysis 40]
Statistical Analysis 78: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 62.2, 95% CI 2-sided [45.9 to 78.4] — [estimate comment as in outcome 6, analysis 40]
Statistical Analysis 79: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — [estimate comment as in outcome 6, analysis 43]
Statistical Analysis 80: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 48.6, 95% CI 2-sided [31.7 to 65.6] — [estimate comment as in outcome 6, analysis 43]
Statistical Analysis 81: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — [estimate comment as in outcome 6, analysis 46]
Statistical Analysis 82: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 51.4, 95% CI 2-sided [34.5 to 68.2] — [estimate comment as in outcome 6, analysis 46]

7. Secondary Outcome: Percentage of Participants With American College of Rheumatology's (ACR) 20/50/70 Response Rates at All Assessment Time Points
Description: The ACR definition for calculating improvement in rheumatoid arthritis is calculated as a 20% improvement (ACR20) in both tender and swollen joint counts and 20% improvement in 3 of the 5 remaining ACR-core set measures: participant and physician global assessments, participant's assessment of arthritis pain, disability, and an acute-phase reactant (i.e. CRP value). Similarly, ACR50 and ACR70 were calculated with the respective percent improvement. The specific components of the ACR assessments are as follows: Tender/Painful Joint count 68 (TJC68), Swollen Joint Count 66 (SJC66), Participant's Assessment of Arthritis Pain, Participant's Global Assessment of Arthritis Disease Activity, Physician's Global Assessment of Arthritis, CRP (mg/L) and Health Assessment Questionnaire - Disability Index (HAQ-DI). For all visits, if any of the component scores were missing, then those scores were considered as not having met the criteria for improvement.
Time Frame: Weeks 1, 2, 4, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and Week 62 (follow-up)
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GSK3196165 22.5 mg | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 135 mg | GSK3196165 180 mg
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37 | 37
Percentage of participants
  Week 1, ACR 20 | 0 | 5 | 8 | 11 | 5 | 19
  Week 1, ACR 50 | 0 | 0 | 3 | 0 | 0 | 0
  Week 1, ACR 70 | 0 | 0 | 0 | 0 | 0 | 0
  Week 2, ACR 20 | 5 | 19 | 14 | 16 | 35 | 43
  Week 2, ACR 50 | 0 | 3 | 3 | 8 | 5 | 5
  Week 2, ACR 70 | 0 | 0 | 0 | 0 | 0 | 0
  Week 4, ACR 20 | 8 | 24 | 35 | 32 | 46 | 46
  Week 4, ACR 50 | 5 | 5 | 5 | 11 | 8 | 8
  Week 4, ACR 70 | 0 | 0 | 0 | 3 | 0 | 5
  Week 6, ACR 20 | 22 | 32 | 30 | 32 | 35 | 46
  Week 6, ACR 50 | 11 | 5 | 8 | 11 | 14 | 14
  Week 6, ACR 70 | 0 | 0 | 3 | 3 | 3 | 5
  Week 8, ACR 20 | 16 | 24 | 41 | 46 | 49 | 51
  Week 8, ACR 50 | 3 | 11 | 14 | 19 | 24 | 19
  Week 8, ACR 70 | 3 | 0 | 3 | 11 | 8 | 8
  Week 12, ACR 20 | 11 | 35 | 41 | 51 | 41 | 51
  Week 12, ACR 50 | 8 | 11 | 27 | 24 | 30 | 22
  Week 12, ACR 70 | 5 | 3 | 14 | 19 | 8 | 11
  Week 16, ACR 20 | 16 | 30 | 46 | 51 | 41 | 68
  Week 16, ACR 50 | 8 | 22 | 27 | 27 | 27 | 22
  Week 16, ACR 70 | 5 | 3 | 14 | 19 | 11 | 11
  Week 20, ACR 20 | 16 | 24 | 38 | 54 | 38 | 59
  Week 20, ACR 50 | 8 | 11 | 24 | 22 | 32 | 30
  Week 20, ACR 70 | 5 | 3 | 16 | 14 | 24 | 19
  Week 24, ACR 20 | 14 | 24 | 41 | 57 | 41 | 59
  Week 24, ACR 50 | 11 | 11 | 27 | 30 | 24 | 27
  Week 24, ACR 70 | 5 | 5 | 14 | 14 | 19 | 19
  Week 28, ACR 20 | 3 | 8 | 19 | 19 | 16 | 68
  Week 28, ACR 50 | 3 | 8 | 16 | 19 | 16 | 24
  Week 28, ACR 70 | 3 | 8 | 14 | 14 | 11 | 14
  Week 32, ACR 20 | 3 | 8 | 22 | 22 | 16 | 54
  Week 32, ACR 50 | 3 | 8 | 22 | 16 | 16 | 30
  Week 32, ACR 70 | 3 | 5 | 19 | 14 | 14 | 16
  Week 36, ACR 20 | 3 | 8 | 19 | 16 | 16 | 59
  Week 36, ACR 50 | 3 | 5 | 19 | 11 | 16 | 35
  Week 36, ACR 70 | 0 | 5 | 19 | 11 | 16 | 14
  Week 40, ACR 20 | 3 | 8 | 19 | 22 | 16 | 54
  Week 40, ACR 50 | 3 | 8 | 16 | 14 | 14 | 32
  Week 40, ACR 70 | 3 | 5 | 16 | 14 | 11 | 16
  Week 44, ACR 20 | 3 | 8 | 19 | 19 | 16 | 54
  Week 44, ACR 50 | 3 | 8 | 19 | 16 | 14 | 38
  Week 44, ACR 70 | 0 | 3 | 19 | 11 | 11 | 19
  Week 48, ACR 20 | 3 | 8 | 19 | 19 | 16 | 57
  Week 48, ACR 50 | 3 | 8 | 19 | 16 | 16 | 35
  Week 48, ACR 70 | 0 | 5 | 19 | 8 | 14 | 22
  Week 52, ACR 20 | 3 | 8 | 16 | 16 | 16 | 51
  Week 52, ACR 50 | 3 | 8 | 16 | 16 | 16 | 27
  Week 52, ACR 70 | 0 | 5 | 16 | 11 | 14 | 14
  Week 62 (follow-up), ACR 20 | 3 | 8 | 16 | 11 | 16 | 43
  Week 62 (follow-up), ACR 50 | 3 | 5 | 16 | 8 | 16 | 27
  Week 62 (follow-up), ACR 70 | 3 | 0 | 16 | 3 | 14 | 19
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — Week 1, ACR20. Difference to Placebo for Week 1 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-0.7 to 16.9] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [0.8 to 20.8] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — Week 1, ACR50. Difference to Placebo for Week 1 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 5: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [-1.1 to 28.1] — Week 2, ACR20. Difference to Placebo for Week 2 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 6: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-5.1 to 21.3] — [estimate comment as in outcome 7, analysis 5]
Statistical Analysis 7: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [-3.1 to 24.7] — [estimate comment as in outcome 7, analysis 5]
Statistical Analysis 8: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — Week 2, ACR50. Difference to Placebo for Week 2 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 9: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — [estimate comment as in outcome 7, analysis 8]
Statistical Analysis 10: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-0.7 to 16.9] — [estimate comment as in outcome 7, analysis 8]
Statistical Analysis 11: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [-0.2 to 32.6] — Week 4, ACR20. Difference to Placebo for Week 4 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 12: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 27.0, 95% CI 2-sided [9.3 to 44.7] — [estimate comment as in outcome 7, analysis 11]
Statistical Analysis 13: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 24.3, 95% CI 2-sided [6.9 to 41.8] — [estimate comment as in outcome 7, analysis 11]
Statistical Analysis 14: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 0.0, 95% CI 2-sided [-10.3 to 10.3] — Week 4, ACR50. Difference to Placebo for Week 4 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 15: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 0.0, 95% CI 2-sided [-10.3 to 10.3] — [estimate comment as in outcome 7, analysis 14]
Statistical Analysis 16: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-7.0 to 17.8] — [estimate comment as in outcome 7, analysis 14]
Statistical Analysis 17: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — Week 4, ACR70. Difference to Placebo for Week 4 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 18: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [-9.3 to 30.9] — Week 6, ACR20. Difference to Placebo for Week 6 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 19: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-11.7 to 27.9] — [estimate comment as in outcome 7, analysis 18]
Statistical Analysis 20: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [-9.3 to 30.9] — [estimate comment as in outcome 7, analysis 18]
Statistical Analysis 21: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = -5.4, 95% CI 2-sided [-17.8 to 7.0] — Week 6, ACR50. Difference to Placebo for Week 6 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 22: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = -2.7, 95% CI 2-sided [-16.0 to 10.6] — [estimate comment as in outcome 7, analysis 21]
Statistical Analysis 23: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 0.0, 95% CI 2-sided [-14.1 to 14.1] — [estimate comment as in outcome 7, analysis 21]
Statistical Analysis 24: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — Week 6, ACR70. Difference to Placebo for Week 6 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 25: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — [estimate comment as in outcome 7, analysis 24]
Statistical Analysis 26: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-10.1 to 26.3] — Week 8, ACR20. Difference to Placebo for Week 8 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 27: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 24.3, 95% CI 2-sided [4.5 to 44.1] — [estimate comment as in outcome 7, analysis 26]
Statistical Analysis 28: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 29.7, 95% CI 2-sided [9.8 to 49.7] — [estimate comment as in outcome 7, analysis 26]
Statistical Analysis 29: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-3.2 to 19.4] — Week 8, ACR50. Difference to Placebo for Week 8 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 30: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [-1.4 to 23.0] — [estimate comment as in outcome 7, analysis 29]
Statistical Analysis 31: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [2.6 to 29.9] — [estimate comment as in outcome 7, analysis 29]
Statistical Analysis 32: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = -2.7, 95% CI 2-sided [-7.9 to 2.5] — Week 8, ACR70. Difference to Placebo for Week 8 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 33: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 0.0, 95% CI 2-sided [-7.4 to 7.4] — [estimate comment as in outcome 7, analysis 32]
Statistical Analysis 34: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-3.2 to 19.4] — [estimate comment as in outcome 7, analysis 32]
Statistical Analysis 35: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 24.3, 95% CI 2-sided [6.0 to 42.7] — Week 12, ACR20. Difference to Placebo for Week 12 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 36: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 29.7, 95% CI 2-sided [11.0 to 48.4] — [estimate comment as in outcome 7, analysis 35]
Statistical Analysis 37: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 40.5, 95% CI 2-sided [21.6 to 59.5] — [estimate comment as in outcome 7, analysis 35]
Statistical Analysis 38: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-10.6 to 16.0] — Week 12, ACR50. Difference to Placebo for Week 12 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 39: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 18.9, 95% CI 2-sided [2.1 to 35.7] — [estimate comment as in outcome 7, analysis 38]
Statistical Analysis 40: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [-0.2 to 32.6] — [estimate comment as in outcome 7, analysis 38]
Statistical Analysis 41: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = -2.7, 95% CI 2-sided [-11.7 to 6.3] — Week 12, ACR70. Difference to Placebo for Week 12 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 42: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-5.1 to 21.3] — [estimate comment as in outcome 7, analysis 41]
Statistical Analysis 43: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [-1.1 to 28.1] — [estimate comment as in outcome 7, analysis 41]
Statistical Analysis 44: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [-5.4 to 32.4] — Week 16, ACR20. Difference to Placebo for Week 16 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 45: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 29.7, 95% CI 2-sided [9.8 to 49.7] — [estimate comment as in outcome 7, analysis 44]
Statistical Analysis 46: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 35.1, 95% CI 2-sided [15.1 to 55.1] — [estimate comment as in outcome 7, analysis 44]
Statistical Analysis 47: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [-2.4 to 29.4] — Week 16, ACR50. Difference to Placebo for Week 16 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 48: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 18.9, 95% CI 2-sided [2.1 to 35.7] — [estimate comment as in outcome 7, analysis 47]
Statistical Analysis 49: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 18.9, 95% CI 2-sided [2.1 to 35.7] — [estimate comment as in outcome 7, analysis 47]
Statistical Analysis 50: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = -2.7, 95% CI 2-sided [-11.7 to 6.3] — Week 16, ACR70. Difference to Placebo for Week 16 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 51: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-5.1 to 21.3] — [estimate comment as in outcome 7, analysis 50]
Statistical Analysis 52: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [-1.1 to 28.1] — [estimate comment as in outcome 7, analysis 50]
Statistical Analysis 53: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-10.1 to 26.3] — Week 20, ACR20. Difference to Placebo for Week 20 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 54: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 21.6, 95% CI 2-sided [2.0 to 41.2] — [estimate comment as in outcome 7, analysis 53]
Statistical Analysis 55: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 37.8, 95% CI 2-sided [17.9 to 57.8] — [estimate comment as in outcome 7, analysis 53]
Statistical Analysis 56: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-10.6 to 16.0] — Week 20, ACR50. Difference to Placebo for Week 20 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 57: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [-0.2 to 32.6] — [estimate comment as in outcome 7, analysis 56]
Statistical Analysis 58: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [-2.4 to 29.4] — [estimate comment as in outcome 7, analysis 56]
Statistical Analysis 59: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = -2.7, 95% CI 2-sided [-11.7 to 6.3] — Week 20, ACR70. Difference to Placebo for Week 20 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 60: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [-3.1 to 24.7] — [estimate comment as in outcome 7, analysis 59]
Statistical Analysis 61: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-5.1 to 21.3] — [estimate comment as in outcome 7, analysis 59]
Statistical Analysis 62: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [-6.9 to 28.5] — Week 24, ACR20. Difference to Placebo for Week 24 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 63: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 27.0, 95% CI 2-sided [7.7 to 46.3] — [estimate comment as in outcome 7, analysis 62]
Statistical Analysis 64: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 43.2, 95% CI 2-sided [23.8 to 62.6] — [estimate comment as in outcome 7, analysis 62]
Statistical Analysis 65: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 0.0, 95% CI 2-sided [-14.1 to 14.1] — Week 24, ACR50. Difference to Placebo for Week 24 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 66: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [-1.2 to 33.7] — [estimate comment as in outcome 7, analysis 65]
Statistical Analysis 67: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 18.9, 95% CI 2-sided [1.1 to 36.7] — [estimate comment as in outcome 7, analysis 65]
Statistical Analysis 68: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 0.0, 95% CI 2-sided [-10.3 to 10.3] — Week 24, ACR70. Difference to Placebo for Week 24 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 69: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-5.1 to 21.3] — [estimate comment as in outcome 7, analysis 68]
Statistical Analysis 70: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-5.1 to 21.3] — [estimate comment as in outcome 7, analysis 68]
Statistical Analysis 71: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-4.8 to 15.6] — Week 28, ACR20. Difference to Placebo for Week 28 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 72: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [2.6 to 29.9] — [estimate comment as in outcome 7, analysis 71]
Statistical Analysis 73: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [2.6 to 29.9] — [estimate comment as in outcome 7, analysis 71]
Statistical Analysis 74: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-4.8 to 15.6] — Week 28, ACR50. Difference to Placebo for Week 28 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 75: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — [estimate comment as in outcome 7, analysis 74]
Statistical Analysis 76: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [2.6 to 29.9] — [estimate comment as in outcome 7, analysis 74]
Statistical Analysis 77: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-4.8 to 15.6] — Week 28, ACR70. Difference to Placebo for Week 28 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 78: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [-1.4 to 23.0] — [estimate comment as in outcome 7, analysis 77]
Statistical Analysis 79: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [-1.4 to 23.0] — [estimate comment as in outcome 7, analysis 77]
Statistical Analysis 80: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-4.8 to 15.6] — Week 32, ACR20. Difference to Placebo for Week 32 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 81: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 18.9, 95% CI 2-sided [4.7 to 33.2] — [estimate comment as in outcome 7, analysis 80]
Statistical Analysis 82: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 18.9, 95% CI 2-sided [4.7 to 33.2] — [estimate comment as in outcome 7, analysis 80]
Statistical Analysis 83: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-4.8 to 15.6] — Week 32, ACR50. Difference to Placebo for Week 32 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 84: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 18.9, 95% CI 2-sided [4.7 to 33.2] — [estimate comment as in outcome 7, analysis 83]
Statistical Analysis 85: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — [estimate comment as in outcome 7, analysis 83]
Statistical Analysis 86: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-6.3 to 11.7] — Week 32, ACR70. Difference to Placebo for Week 32 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 87: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [2.6 to 29.9] — [estimate comment as in outcome 7, analysis 86]
Statistical Analysis 88: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [-1.4 to 23.0] — [estimate comment as in outcome 7, analysis 86]
Statistical Analysis 89: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-4.8 to 15.6] — Week 36, ACR20. Difference to Placebo for Week 36 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 90: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [2.6 to 29.9] — [estimate comment as in outcome 7, analysis 89]
Statistical Analysis 91: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — [estimate comment as in outcome 7, analysis 89]
Statistical Analysis 92: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-6.3 to 11.7] — Week 36, ACR50. Difference to Placebo for Week 36 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 93: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [2.6 to 29.9] — [estimate comment as in outcome 7, analysis 92]
Statistical Analysis 94: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-3.2 to 19.4] — [estimate comment as in outcome 7, analysis 92]
Statistical Analysis 95: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — Week 36, ACR70. Difference to Placebo for Week 36 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 96: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 18.9, 95% CI 2-sided [6.3 to 31.5] — [estimate comment as in outcome 7, analysis 95]
Statistical Analysis 97: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [0.8 to 20.8] — [estimate comment as in outcome 7, analysis 95]
Statistical Analysis 98: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-4.8 to 15.6] — Week 40, ACR20. Difference to Placebo for Week 40 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 99: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [2.6 to 29.9] — [estimate comment as in outcome 7, analysis 98]
Statistical Analysis 100: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 18.9, 95% CI 2-sided [4.7 to 33.2] — [estimate comment as in outcome 7, analysis 98]
Statistical Analysis 101: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-4.8 to 15.6] — Week 40, ACR50. Difference to Placebo for Week 40 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 102: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — [estimate comment as in outcome 7, analysis 101]
Statistical Analysis 103: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [-1.4 to 23.0] — [estimate comment as in outcome 7, analysis 101]
Statistical Analysis 104: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-6.3 to 11.7] — Week 40, ACR70. Difference to Placebo for Week 40 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 105: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — [estimate comment as in outcome 7, analysis 104]
Statistical Analysis 106: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [-1.4 to 23.0] — [estimate comment as in outcome 7, analysis 104]
Statistical Analysis 107: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-4.8 to 15.6] — Week 44, ACR20. Difference to Placebo for Week 44 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 108: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [2.6 to 29.9] — [estimate comment as in outcome 7, analysis 107]
Statistical Analysis 109: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [2.6 to 29.9] — [estimate comment as in outcome 7, analysis 107]
Statistical Analysis 110: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-4.8 to 15.6] — Week 44, ACR50. Difference to Placebo for Week 44 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 111: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [2.6 to 29.9] — [estimate comment as in outcome 7, analysis 110]
Statistical Analysis 112: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — [estimate comment as in outcome 7, analysis 110]
Statistical Analysis 113: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — Week 44, ACR70. Difference to Placebo for Week 44 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 114: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 18.9, 95% CI 2-sided [6.3 to 31.5] — [estimate comment as in outcome 7, analysis 113]
Statistical Analysis 115: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [0.8 to 20.8] — [estimate comment as in outcome 7, analysis 113]
Statistical Analysis 116: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-4.8 to 15.6] — Week 48, ACR20. Difference to Placebo for Week 48 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 117: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [2.6 to 29.9] — [estimate comment as in outcome 7, analysis 116]
Statistical Analysis 118: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [2.6 to 29.9] — [estimate comment as in outcome 7, analysis 116]
Statistical Analysis 119: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — Week 48, ACR50. Difference to Placebo for Week 48 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 120: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [2.6 to 29.9] — [estimate comment as in outcome 7, analysis 119]
Statistical Analysis 121: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [2.6 to 29.9] — [estimate comment as in outcome 7, analysis 119]
Statistical Analysis 122: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — Week 48, ACR70. Difference to Placebo for Week 48 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 123: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 18.9, 95% CI 2-sided [6.3 to 31.5] — [estimate comment as in outcome 7, analysis 122]
Statistical Analysis 124: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-0.7 to 16.9] — [estimate comment as in outcome 7, analysis 122]
Statistical Analysis 125: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-4.8 to 15.6] — Week 52, ACR20. Difference to Placebo for Week 52 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 126: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — [estimate comment as in outcome 7, analysis 125]
Statistical Analysis 127: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — [estimate comment as in outcome 7, analysis 125]
Statistical Analysis 128: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-4.8 to 15.6] — Week 52, ACR50. Difference to Placebo for Week 52 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 129: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — [estimate comment as in outcome 7, analysis 128]
Statistical Analysis 130: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — [estimate comment as in outcome 7, analysis 128]
Statistical Analysis 131: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — Week 52, ACR70. Difference to Placebo for Week 52 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 132: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [4.3 to 28.1] — [estimate comment as in outcome 7, analysis 131]
Statistical Analysis 133: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [0.8 to 20.8] — [estimate comment as in outcome 7, analysis 131]
Statistical Analysis 134: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-4.8 to 15.6] — Week 62 (follow-up), ACR20. Difference to Placebo for Week 62 (follow-up) is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 135: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — [estimate comment as in outcome 7, analysis 134]
Statistical Analysis 136: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-3.2 to 19.4] — [estimate comment as in outcome 7, analysis 134]
Statistical Analysis 137: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-6.3 to 11.7] — Week 62 (follow-up), ACR50. Difference to Placebo for Week 62 (follow-up) is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 138: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — [estimate comment as in outcome 7, analysis 137]
Statistical Analysis 139: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-4.8 to 15.6] — [estimate comment as in outcome 7, analysis 137]
Statistical Analysis 140: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = -2.7, 95% CI 2-sided [-7.9 to 2.5] — Week 62 (follow-up), ACR70. Difference to Placebo for Week 62 (follow-up) is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 141: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — [estimate comment as in outcome 7, analysis 140]
Statistical Analysis 142: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 0.0, 95% CI 2-sided [-7.4 to 7.4] — [estimate comment as in outcome 7, analysis 140]
Statistical Analysis 143: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — Week 1, ACR20. Difference to Placebo is presented for Week 1. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 144: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 18.9, 95% CI 2-sided [6.3 to 31.5] — [estimate comment as in outcome 7, analysis 143]
Statistical Analysis 145: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 29.7, 95% CI 2-sided [12.7 to 46.8] — Week 2, ACR20. Difference to Placebo is presented for Week 2. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 146: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 37.8, 95% CI 2-sided [20.3 to 55.4] — [estimate comment as in outcome 7, analysis 145]
Statistical Analysis 147: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — Week 2, ACR50. Difference to Placebo is presented for Week 2. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 148: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 7, analysis 147]
Statistical Analysis 149: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 37.8, 95% CI 2-sided [19.5 to 56.1] — Week 4, ACR20. Difference to Placebo is presented for Week 4. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 150: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 51.4, 95% CI 2-sided [19.5 to 56.1] — [estimate comment as in outcome 7, analysis 149]
Statistical Analysis 151: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-8.7 to 14.1] — Week 4, ACR50. Difference to Placebo is presented for Week 4. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 152: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-8.7 to 14.1] — [estimate comment as in outcome 7, analysis 151]
Statistical Analysis 153: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — Week 4, ACR70. Difference to Placebo is presented for Week 4. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 154: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [-6.8 to 33.8] — Week 6, ACR20. Difference to Placebo is presented for Week 6. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 155: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 24.3, 95% CI 2-sided [3.5 to 45.2] — [estimate comment as in outcome 7, analysis 154]
Statistical Analysis 156: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-12.2 to 17.6] — Week 6, ACR50. Difference to Placebo is presented for Week 6. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 157: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-12.2 to 17.6] — [estimate comment as in outcome 7, analysis 156]
Statistical Analysis 158: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — Week 6, ACR70. Difference to Placebo is presented for Week 6. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 159: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 7, analysis 158]
Statistical Analysis 160: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 32.4, 95% CI 2-sided [12.4 to 52.4] — Week 8, ACR20. Difference to Placebo is presented for Week 8. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 161: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 35.1, 95% CI 2-sided [15.1 to 55.1] — [estimate comment as in outcome 7, analysis 160]
Statistical Analysis 162: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 21.6, 95% CI 2-sided [6.8 to 36.4] — Week 8, ACR50. Difference to Placebo is presented for Week 8. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 163: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [2.6 to 29.9] — [estimate comment as in outcome 7, analysis 162]
Statistical Analysis 164: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-4.8 to 15.6] — Week 8, ACR70. Difference to Placebo is presented for Week 8. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 165: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-4.8 to 15.6] — [estimate comment as in outcome 7, analysis 164]
Statistical Analysis 166: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 29.7, 95% CI 2-sided [11.0 to 48.4] — Week 12, ACR20. Difference to Placebo is presented for Week 8. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 167: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 40.5, 95% CI 2-sided [21.6 to 59.5] — [estimate comment as in outcome 7, analysis 166]
Statistical Analysis 168: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 21.6, 95% CI 2-sided [4.5 to 38.8] — Week 12, ACR50. Difference to Placebo is presented for Week 12. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 169: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [-2.4 to 29.4] — [estimate comment as in outcome 7, analysis 168]
Statistical Analysis 170: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-8.7 to 14.1] — Week 12, ACR70. Difference to Placebo is presented for Week 12. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 171: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-7.0 to 17.8] — [estimate comment as in outcome 7, analysis 170]
Statistical Analysis 172: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 24.3, 95% CI 2-sided [4.5 to 44.1] — Week 16, ACR20. Difference to Placebo is presented for Week 16. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 173: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 51.4, 95% CI 2-sided [32.2 to 70.5] — [estimate comment as in outcome 7, analysis 172]
Statistical Analysis 174: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 18.9, 95% CI 2-sided [2.1 to 35.7] — Week 16, ACR50. Difference to Placebo is presented for Week 16. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 175: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [-2.4 to 29.4] — [estimate comment as in outcome 7, analysis 174]
Statistical Analysis 176: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-7.0 to 17.8] — Week 16, ACR70. Difference to Placebo is presented for Week 16. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 177: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 21.6, 95% CI 2-sided [2.0 to 41.2] — Week 20, ACR20. Difference to Placebo is presented for Week 20. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 178: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 43.2, 95% CI 2-sided [23.5 to 63.0] — [estimate comment as in outcome 7, analysis 177]
Statistical Analysis 179: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 24.3, 95% CI 2-sided [6.9 to 41.8] — Week 20, ACR50. Difference to Placebo is presented for Week 20. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 180: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 21.6, 95% CI 2-sided [4.5 to 38.8] — [estimate comment as in outcome 7, analysis 179]
Statistical Analysis 181: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 18.9, 95% CI 2-sided [3.3 to 34.5] — Week 20, ACR70. Difference to Placebo is presented for Week 20. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 182: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [-1.1 to 28.1] — [estimate comment as in outcome 7, analysis 181]
Statistical Analysis 183: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 27.0, 95% CI 2-sided [7.7 to 46.3] — Week 24, ACR20. Difference to Placebo is presented for Week 24. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 184: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 45.9, 95% CI 2-sided [26.7 to 65.2] — [estimate comment as in outcome 7, analysis 183]
Statistical Analysis 185: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [-3.6 to 30.6] — Week 24, ACR50. Difference to Placebo is presented for Week 24. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 186: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [-1.2 to 33.7] — [estimate comment as in outcome 7, analysis 185]
Statistical Analysis 187: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [-1.1 to 28.1] — Week 24, ACR70. Difference to Placebo is presented for Week 24. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 188: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [-1.1 to 28.1] — [estimate comment as in outcome 7, analysis 187]
Statistical Analysis 189: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — Week 28, ACR20. Difference to Placebo is presented for Week 28. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 190: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 64.9, 95% CI 2-sided [48.9 to 80.8] — [estimate comment as in outcome 7, analysis 189]
Statistical Analysis 191: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — Week 28, ACR50. Difference to Placebo is presented for Week 28. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 192: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 21.6, 95% CI 2-sided [6.8 to 36.4] — [estimate comment as in outcome 7, analysis 191]
Statistical Analysis 193: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-3.2 to 19.4] — Week 28, ACR70. Difference to Placebo is presented for Week 28. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 194: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [-1.4 to 23.0] — [estimate comment as in outcome 7, analysis 193]
Statistical Analysis 195: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — Week 32, ACR20. Difference to Placebo is presented for Week 32. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 196: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 51.4, 95% CI 2-sided [34.5 to 68.2] — [estimate comment as in outcome 7, analysis 195]
Statistical Analysis 197: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — Week 32, ACR50. Difference to Placebo is presented for Week 32. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 198: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 27.0, 95% CI 2-sided [11.4 to 42.7] — [estimate comment as in outcome 7, analysis 197]
Statistical Analysis 199: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [-1.4 to 23.0] — Week 32, ACR70. Difference to Placebo is presented for Week 32. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 200: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — [estimate comment as in outcome 7, analysis 199]
Statistical Analysis 201: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — Week 36, ACR20. Difference to Placebo is presented for Week 36. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 202: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 56.8, 95% CI 2-sided [40.1 to 73.4] — [estimate comment as in outcome 7, analysis 201]
Statistical Analysis 203: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — Week 36, ACR50. Difference to Placebo is presented for Week 36. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 204: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 32.4, 95% CI 2-sided [16.2 to 48.7] — [estimate comment as in outcome 7, analysis 203]
Statistical Analysis 205: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [4.3 to 28.1] — Week 36, ACR70. Difference to Placebo is presented for Week 36. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 206: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [2.5 to 24.5] — [estimate comment as in outcome 7, analysis 205]
Statistical Analysis 207: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — Week 40, ACR20. Difference to Placebo is presented for Week 40. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 208: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 51.4, 95% CI 2-sided [34.5 to 68.2] — [estimate comment as in outcome 7, analysis 207]
Statistical Analysis 209: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [-1.4 to 23.0] — Week 40, ACR50. Difference to Placebo is presented for Week 40. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 210: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 29.7, 95% CI 2-sided [13.8 to 45.7] — [estimate comment as in outcome 7, analysis 209]
Statistical Analysis 211: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-3.2 to 19.4] — Week 40, ACR70. Difference to Placebo is presented for Week 40. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 212: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — [estimate comment as in outcome 7, analysis 211]
Statistical Analysis 213: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — Week 44, ACR20. Difference to Placebo is presented for Week 44. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 214: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 51.4, 95% CI 2-sided [34.5 to 68.2] — [estimate comment as in outcome 7, analysis 213]
Statistical Analysis 215: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [-1.4 to 23.0] — Week 44, ACR50. Difference to Placebo is presented for Week 44. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 216: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 35.1, 95% CI 2-sided [18.7 to 51.6] — [estimate comment as in outcome 7, analysis 215]
Statistical Analysis 217: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [0.8 to 20.8] — Week 44, ACR70. Difference to Placebo is presented for Week 44. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 218: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 18.9, 95% CI 2-sided [6.3 to 31.5] — [estimate comment as in outcome 7, analysis 217]
Statistical Analysis 219: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — Week 48, ACR20. Difference to Placebo is presented for Week 48. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 220: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 51.4, 95% CI 2-sided [37.3 to 70.9] — [estimate comment as in outcome 7, analysis 219]
Statistical Analysis 221: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — Week 48, ACR50. Difference to Placebo is presented for Week 48. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 222: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 32.4, 95% CI 2-sided [16.2 to 48.7] — [estimate comment as in outcome 7, analysis 221]
Statistical Analysis 223: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [2.5 to 24.5] — Week 48, ACR70. Difference to Placebo is presented for Week 48. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 224: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 21.6, 95% CI 2-sided [8.4 to 34.9] — [estimate comment as in outcome 7, analysis 223]
Statistical Analysis 225: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — Week 52, ACR20. Difference to Placebo is presented for Week 52. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 226: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 48.6, 95% CI 2-sided [31.7 to 65.6] — [estimate comment as in outcome 7, analysis 225]
Statistical Analysis 227: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — Week 52, ACR50. Difference to Placebo is presented for Week 52. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 228: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 24.3, 95% CI 2-sided [9.1 to 39.6] — [estimate comment as in outcome 7, analysis 227]
Statistical Analysis 229: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [2.5 to 24.5] — Week 52, ACR70. Difference to Placebo is presented for Week 52. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 230: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [2.5 to 24.5] — [estimate comment as in outcome 7, analysis 229]
Statistical Analysis 231: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — Week 62 (follow-up), ACR20. Difference to Placebo is presented for Week 62 (follow-up). 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 232: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 40.5, 95% CI 2-sided [23.7 to 57.3] — [estimate comment as in outcome 7, analysis 231]
Statistical Analysis 233: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [0.5 to 26.5] — Week 62 (follow-up), ACR50. Difference to Placebo is presented for Week 62 (follow-up). 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 234: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 24.3, 95% CI 2-sided [9.1 to 39.6] — [estimate comment as in outcome 7, analysis 233]
Statistical Analysis 235: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [-1.4 to 23.0] — Week 62 (follow-up), ACR70. Difference to Placebo is presented for Week 62 (follow-up). 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 236: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [2.6 to 29.9] — [estimate comment as in outcome 7, analysis 235]

8. Secondary Outcome: Percentage of Participants With Index-based ACR/EULAR Remission Rates at All Assessment Time Points
Description: Index-based remission was achieved if the following requirement was met: SDAI <= 3.3. If the SDAI value was missing at an individual assessment point, Index-based remission for that assessment was set to missing.
Time Frame: Weeks 1, 2, 4, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and Week 62 (follow-up)
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GSK3196165 22.5 mg | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 135 mg | GSK3196165 180 mg
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37 | 37
Percentage of participants
  Index based ACR/EULAR, Week 1 | 0 | 0 | 0 | 0 | 0 | 0
  Index based ACR/EULAR, Week 2 | 0 | 0 | 0 | 0 | 0 | 3
  Index based ACR/EULAR, Week 4 | 0 | 0 | 0 | 3 | 0 | 3
  Index based ACR/EULAR, Week 6 | 0 | 0 | 0 | 3 | 3 | 3
  Index based ACR/EULAR, Week 8 | 3 | 0 | 0 | 3 | 3 | 3
  Index based ACR/EULAR, Week 12 | 3 | 0 | 0 | 3 | 3 | 3
  Index based ACR/EULAR, Week 16 | 0 | 0 | 3 | 14 | 3 | 5
  Index based ACR/EULAR, Week 20 | 0 | 0 | 5 | 11 | 3 | 5
  Index based ACR/EULAR, Week 24 | 0 | 0 | 5 | 8 | 8 | 5
  Index based ACR/EULAR, Week 28 | 0 | 0 | 5 | 11 | 8 | 14
  Index based ACR/EULAR, Week 32 | 0 | 0 | 14 | 8 | 8 | 11
  Index based ACR/EULAR, Week 36 | 0 | 3 | 11 | 8 | 14 | 5
  Index based ACR/EULAR, Week 40 | 0 | 3 | 11 | 8 | 5 | 14
  Index based ACR/EULAR, Week 44 | 0 | 3 | 8 | 11 | 5 | 8
  Index based ACR/EULAR, Week 48 | 0 | 3 | 11 | 8 | 11 | 3
  Index based ACR/EULAR, Week 52 | 0 | 5 | 14 | 5 | 5 | 8
  Index based ACR/EULAR, Week 62 (follow-up) | 0 | 0 | 8 | 3 | 5 | 14
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — Index based ACR/EULAR, Week 4. Difference to Placebo for Week 4 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — Index based ACR/EULAR, Week 6. Difference to Placebo for Week 6 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = -2.7, 95% CI 2-sided [-7.9 to 2.5] — Index based ACR/EULAR, Week 8. Difference to Placebo for Week 8 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = -2.7, 95% CI 2-sided [-7.9 to 2.5] — [estimate comment as in outcome 8, analysis 3]
Statistical Analysis 5: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 0.0, 95% CI 2-sided [-7.4 to 7.4] — [estimate comment as in outcome 8, analysis 3]
Statistical Analysis 6: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = -2.7, 95% CI 2-sided [-7.9 to 2.5] — Index based ACR/EULAR, Week 12. Difference to Placebo for Week 12 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 7: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = -2.7, 95% CI 2-sided [-7.9 to 2.5] — [estimate comment as in outcome 8, analysis 6]
Statistical Analysis 8: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 0.0, 95% CI 2-sided [-7.4 to 7.4] — [estimate comment as in outcome 8, analysis 6]
Statistical Analysis 9: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — Index based ACR/EULAR, Week 16. Difference to Placebo for Week 16 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 10: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [2.5 to 24.5] — [estimate comment as in outcome 8, analysis 9]
Statistical Analysis 11: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — Index based ACR/EULAR, Week 20. Difference to Placebo for Week 20 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 12: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [0.8 to 20.8] — [estimate comment as in outcome 8, analysis 11]
Statistical Analysis 13: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — Index based ACR/EULAR, Week 24. Difference to Placebo for Week 24 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 14: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-0.7 to 16.9] — [estimate comment as in outcome 8, analysis 13]
Statistical Analysis 15: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — Index based ACR/EULAR, Week 28. Difference to Placebo for Week 28 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 16: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [0.8 to 20.8] — [estimate comment as in outcome 8, analysis 15]
Statistical Analysis 17: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [2.5 to 24.5] — Index based ACR/EULAR, Week 32. Difference to Placebo for Week 32 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 18: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-0.7 to 16.9] — [estimate comment as in outcome 8, analysis 17]
Statistical Analysis 19: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — Index based ACR/EULAR, Week 36. Difference to Placebo for Week 36 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 20: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [0.8 to 20.8] — [estimate comment as in outcome 8, analysis 19]
Statistical Analysis 21: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-0.7 to 16.9] — [estimate comment as in outcome 8, analysis 19]
Statistical Analysis 22: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — Index based ACR/EULAR, Week 40. Difference to Placebo for Week 40 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 23: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [0.8 to 20.8] — [estimate comment as in outcome 8, analysis 22]
Statistical Analysis 24: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-0.7 to 16.9] — [estimate comment as in outcome 8, analysis 22]
Statistical Analysis 25: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — Index based ACR/EULAR, Week 44. Difference to Placebo for Week 44 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 26: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-0.7 to 16.9] — [estimate comment as in outcome 8, analysis 25]
Statistical Analysis 27: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [0.8 to 20.8] — [estimate comment as in outcome 8, analysis 25]
Statistical Analysis 28: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — Index based ACR/EULAR, Week 48. Difference to Placebo for Week 48 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 29: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [0.8 to 20.8] — [estimate comment as in outcome 8, analysis 28]
Statistical Analysis 30: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-0.7 to 16.9] — [estimate comment as in outcome 8, analysis 28]
Statistical Analysis 31: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — Index based ACR/EULAR, Week 52. Difference to Placebo for Week 52 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 32: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [2.5 to 24.5] — [estimate comment as in outcome 8, analysis 31]
Statistical Analysis 33: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 8, analysis 31]
Statistical Analysis 34: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-0.7 to 16.9] — Index based ACR/EULAR, Week 62 (follow-up). Difference to Placebo for Week 62 (follow-up) is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 35: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — [estimate comment as in outcome 8, analysis 34]
Statistical Analysis 36: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — Index based ACR/EULAR, Week 2. Difference to Placebo for Week 2 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 37: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 38: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — [estimate comment as in outcome 8, analysis 2]
Statistical Analysis 39: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — [estimate comment as in outcome 8, analysis 2]
Statistical Analysis 40: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 0.0, 95% CI 2-sided [-7.4 to 7.4] — [estimate comment as in outcome 8, analysis 3]
Statistical Analysis 41: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 0.0, 95% CI 2-sided [-7.4 to 7.4] — [estimate comment as in outcome 8, analysis 3]
Statistical Analysis 42: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 0.0, 95% CI 2-sided [-7.4 to 7.4] — [estimate comment as in outcome 8, analysis 6]
Statistical Analysis 43: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 0.0, 95% CI 2-sided [-7.4 to 7.4] — [estimate comment as in outcome 8, analysis 6]
Statistical Analysis 44: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — [estimate comment as in outcome 8, analysis 9]
Statistical Analysis 45: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 8, analysis 9]
Statistical Analysis 46: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 12.7] — [estimate comment as in outcome 8, analysis 11]
Statistical Analysis 47: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 68.2] — [estimate comment as in outcome 8, analysis 11]
Statistical Analysis 48: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-0.7 to 16.9] — [estimate comment as in outcome 8, analysis 13]
Statistical Analysis 49: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 8, analysis 13]
Statistical Analysis 50: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-0.7 to 16.9] — [estimate comment as in outcome 8, analysis 15]
Statistical Analysis 51: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [2.5 to 24.5] — [estimate comment as in outcome 8, analysis 15]
Statistical Analysis 52: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-0.7 to 16.9] — [estimate comment as in outcome 8, analysis 17]
Statistical Analysis 53: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [0.8 to 20.8] — [estimate comment as in outcome 8, analysis 17]
Statistical Analysis 54: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [2.5 to 24.5] — [estimate comment as in outcome 8, analysis 19]
Statistical Analysis 55: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 8, analysis 19]
Statistical Analysis 56: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 8, analysis 22]
Statistical Analysis 57: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [2.5 to 24.5] — [estimate comment as in outcome 8, analysis 22]
Statistical Analysis 58: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 8, analysis 25]
Statistical Analysis 59: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-0.7 to 16.9] — [estimate comment as in outcome 8, analysis 25]
Statistical Analysis 60: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [0.8 to 20.8] — [estimate comment as in outcome 8, analysis 28]
Statistical Analysis 61: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — [estimate comment as in outcome 8, analysis 28]
Statistical Analysis 62: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 8, analysis 31]
Statistical Analysis 63: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-0.7 to 16.9] — [estimate comment as in outcome 8, analysis 31]
Statistical Analysis 64: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 8, analysis 34]
Statistical Analysis 65: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [2.5 to 24.5] — [estimate comment as in outcome 8, analysis 34]

9. Secondary Outcome: Percentage of Participants With Boolean-based ACR/EULAR Remission Rates at All Assessment Time Points
Description: Boolean-based remission was achieved if all of the following requirements were met at the same time: TJC68 <= 1,SJC66 <= 1,CRP <= 1mg/dL, PtGA <= 10. If one of the components was missing at an individual assessment point, Boolean-based remission for that assessment was set to missing.
Time Frame: Weeks 1, 2, 4, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and Week 62 (follow-up)
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GSK3196165 22.5 mg | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 135 mg | GSK3196165 180 mg
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37 | 37
Percentage of participants
  Boolean based ACR/EULAR, Week 1 | 0 | 0 | 0 | 0 | 0 | 0
  Boolean based ACR/EULAR, Week 2 | 0 | 0 | 0 | 0 | 0 | 3
  Boolean based ACR/EULAR, Week 4 | 0 | 0 | 0 | 0 | 0 | 0
  Boolean based ACR/EULAR, Week 6 | 0 | 0 | 0 | 0 | 3 | 3
  Boolean based ACR/EULAR, Week 8 | 0 | 0 | 0 | 3 | 3 | 5
  Boolean based ACR/EULAR, Week 12 | 0 | 0 | 0 | 8 | 0 | 3
  Boolean based ACR/EULAR, Week 16 | 0 | 0 | 3 | 5 | 3 | 5
  Boolean based ACR/EULAR, Week 20 | 0 | 0 | 5 | 8 | 3 | 5
  Boolean based ACR/EULAR, Week 24 | 0 | 0 | 3 | 8 | 5 | 3
  Boolean based ACR/EULAR, Week 28 | 0 | 0 | 5 | 8 | 5 | 5
  Boolean based ACR/EULAR, Week 32 | 0 | 0 | 5 | 5 | 5 | 5
  Boolean based ACR/EULAR, Week 36 | 0 | 0 | 8 | 5 | 8 | 3
  Boolean based ACR/EULAR, Week 40 | 0 | 0 | 8 | 8 | 5 | 8
  Boolean based ACR/EULAR, Week 44 | 0 | 0 | 11 | 8 | 5 | 5
  Boolean based ACR/EULAR, Week 48 | 0 | 3 | 8 | 3 | 11 | 3
  Boolean based ACR/EULAR, Week 52 | 0 | 0 | 11 | 3 | 5 | 5
  Boolean based ACR/EULAR, Week 62 (follow-up) | 0 | 0 | 8 | 3 | 3 | 5
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — Boolean based ACR/EULAR, Week 8. Difference to Placebo for Week 8 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-0.7 to 16.9] — Boolean based ACR/EULAR, Week 12. Difference to Placebo for Week 12 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — [estimate comment as in outcome 6, analysis 19]
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — Boolean based ACR/EULAR, Week 16. Difference to Placebo for Week 16 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 5: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — Boolean based ACR/EULAR, Week 20. Difference to Placebo for Week 20 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 6: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-0.7 to 16.9] — [estimate comment as in outcome 9, analysis 5]
Statistical Analysis 7: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — Boolean based ACR/EULAR, Week 24. Difference to Placebo for Week 24 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 8: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-0.7 to 16.9] — [estimate comment as in outcome 9, analysis 7]
Statistical Analysis 9: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — Boolean based ACR/EULAR, Week 28. Difference to Placebo for Week 28 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 10: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-0.7 to 16.9] — [estimate comment as in outcome 9, analysis 9]
Statistical Analysis 11: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — Boolean based ACR/EULAR, Week 32. Difference to Placebo for Week 32 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 12: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 9, analysis 11]
Statistical Analysis 13: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-0.7 to 16.9] — Boolean based ACR/EULAR, Week 36. Difference to Placebo for Week 36 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 14: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 9, analysis 13]
Statistical Analysis 15: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-0.7 to 16.9] — Boolean based ACR/EULAR, Week 40. Difference to Placebo for Week 40 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 16: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-0.7 to 16.9] — [estimate comment as in outcome 9, analysis 15]
Statistical Analysis 17: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [0.8 to 20.8] — Boolean based ACR/EULAR, Week 44. Difference to Placebo for Week 44 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 18: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-0.7 to 16.9] — [estimate comment as in outcome 9, analysis 17]
Statistical Analysis 19: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — Boolean based ACR/EULAR, Week 48. Difference to Placebo for Week 48 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 20: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — [estimate comment as in outcome 9, analysis 19]
Statistical Analysis 21: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 21.6, 95% CI 2-sided [0.4 to 42.8] — [estimate comment as in outcome 9, analysis 19]
Statistical Analysis 22: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [0.8 to 20.8] — Boolean based ACR/EULAR, Week 52. Difference to Placebo for Week 52 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 23: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — [estimate comment as in outcome 9, analysis 22]
Statistical Analysis 24: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-0.7 to 16.9] — Boolean based ACR/EULAR, Week 62 (follow-up). Difference to Placebo for Week 62 (follow-up) is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 25: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — [estimate comment as in outcome 9, analysis 24]
Statistical Analysis 26: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — Boolean based ACR/EULAR, Week 2. Difference to Placebo for Week 2 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 27: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — Boolean based ACR/EULAR, Week 6. Difference to Placebo for Week 6 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 28: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — [estimate comment as in outcome 9, analysis 27]
Statistical Analysis 29: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 30: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 31: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — [estimate comment as in outcome 9, analysis 2]
Statistical Analysis 32: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — [estimate comment as in outcome 9, analysis 4]
Statistical Analysis 33: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 9, analysis 4]
Statistical Analysis 34: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — [estimate comment as in outcome 9, analysis 5]
Statistical Analysis 35: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 9, analysis 5]
Statistical Analysis 36: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 9, analysis 7]
Statistical Analysis 37: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — [estimate comment as in outcome 9, analysis 7]
Statistical Analysis 38: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 9, analysis 9]
Statistical Analysis 39: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 9, analysis 9]
Statistical Analysis 40: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 9, analysis 11]
Statistical Analysis 41: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 9, analysis 11]
Statistical Analysis 42: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-0.7 to 16.9] — [estimate comment as in outcome 9, analysis 13]
Statistical Analysis 43: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — [estimate comment as in outcome 9, analysis 13]
Statistical Analysis 44: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 9, analysis 15]
Statistical Analysis 45: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-0.7 to 16.9] — [estimate comment as in outcome 9, analysis 15]
Statistical Analysis 46: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 9, analysis 17]
Statistical Analysis 47: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 9, analysis 17]
Statistical Analysis 48: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [0.8 to 20.8] — [estimate comment as in outcome 9, analysis 19]
Statistical Analysis 49: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — [estimate comment as in outcome 9, analysis 19]
Statistical Analysis 50: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 9, analysis 22]
Statistical Analysis 51: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 9, analysis 22]
Statistical Analysis 52: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — [estimate comment as in outcome 9, analysis 24]
Statistical Analysis 53: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 9, analysis 24]

10. Secondary Outcome: Percentage of Participants in Clinical Disease Activity Index (CDAI) Remission
Description: CDAI combines information relating to the number of swollen and tender joints, in addition to a measure of general health from both the participants and the physician. CDAI utilizing joint scores from the following 28 joints: elbows, shoulders, elbow, wrists, metacarpal- phalangeal I-V, proximal interphalangeal I-V and knees and is calculated using the following formula: CDAI =TJC28 + SJC28 + GH + GP Where TJC - Tender joint Count, SJC= Swollen Joint Count, (GH=participant assessment of disease activity and GP=physician assessment of disease activity using a 10 cm visual analogue scale with 0 = best, 100 = worst). It ranges between 0 and 76. High score indicates worse outcome, low score indicates better outcome. Remission was achieved for a non-missing CDAI value <=2.8.
Time Frame: Weeks 1, 2, 4, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and Week 62 (follow-up)
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GSK3196165 22.5 mg | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 135 mg | GSK3196165 180 mg
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37 | 37
Percentage of participants
  CDAI, Week 1 | 0 | 0 | 0 | 0 | 0 | 0
  CDAI, Week 2 | 0 | 0 | 0 | 0 | 0 | 5
  CDAI, Week 4 | 0 | 0 | 0 | 5 | 0 | 3
  CDAI, Week 6 | 0 | 0 | 0 | 3 | 3 | 3
  CDAI, Week 8 | 3 | 0 | 0 | 3 | 3 | 3
  CDAI, Week 12 | 3 | 0 | 0 | 11 | 3 | 5
  CDAI, Week 16 | 0 | 3 | 3 | 16 | 3 | 5
  CDAI, Week 20 | 0 | 0 | 3 | 11 | 3 | 5
  CDAI, Week 24 | 0 | 0 | 5 | 5 | 8 | 5
  CDAI, Week 28 | 0 | 0 | 3 | 11 | 5 | 14
  CDAI, Week 32 | 0 | 0 | 14 | 8 | 8 | 11
  CDAI, Week 36 | 0 | 3 | 11 | 8 | 14 | 5
  CDAI, Week 40 | 0 | 3 | 11 | 8 | 5 | 14
  CDAI, Week 44 | 0 | 3 | 11 | 11 | 5 | 5
  CDAI, Week 48 | 0 | 3 | 14 | 8 | 11 | 8
  CDAI, Week 52 | 0 | 0 | 14 | 5 | 5 | 8
  CDAI, Week 62 (follow-up) | 0 | 0 | 8 | 3 | 5 | 16
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — CDAI, Week 4, Difference to Placebo for Week 4 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — CDAI, Week 6. Difference to Placebo for Week 6 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = -2.7, 95% CI 2-sided [-7.9 to 2.5] — CDAI, Week 8. Difference to Placebo for Week 8 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = -2.7, 95% CI 2-sided [-7.9 to 2.5] — [estimate comment as in outcome 10, analysis 3]
Statistical Analysis 5: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 0.0, 95% CI 2-sided [-7.4 to 7.4] — [estimate comment as in outcome 10, analysis 3]
Statistical Analysis 6: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = -2.7, 95% CI 2-sided [-7.9 to 2.5] — CDAI, Week 12. Difference to Placebo for Week 12 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 7: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = -2.7, 95% CI 2-sided [-7.9 to 2.5] — [estimate comment as in outcome 10, analysis 6]
Statistical Analysis 8: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-3.2 to 19.4] — [estimate comment as in outcome 10, analysis 6]
Statistical Analysis 9: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — CDAI, Week 16. Difference to Placebo for Week 16 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 10: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — [estimate comment as in outcome 10, analysis 9]
Statistical Analysis 11: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [4.3 to 28.1] — [estimate comment as in outcome 10, analysis 9]
Statistical Analysis 12: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — CDAI, Week 20. Difference to Placebo for Week 20 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 13: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [0.8 to 20.8] — [estimate comment as in outcome 10, analysis 12]
Statistical Analysis 14: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — CDAI, Week 24. Difference to Placebo for Week 24 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 15: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 10, analysis 14]
Statistical Analysis 16: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — CDAI, Week 28. Difference to Placebo for Week 28 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 17: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [0.8 to 20.8] — [estimate comment as in outcome 10, analysis 16]
Statistical Analysis 18: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [2.5 to 24.5] — CDAI, Week 32. Difference to Placebo for Week 32 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 19: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-0.7 to 16.9] — [estimate comment as in outcome 10, analysis 18]
Statistical Analysis 20: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — CDAI, Week 36. Difference to Placebo for Week 36 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 21: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [0.8 to 20.8] — [estimate comment as in outcome 10, analysis 20]
Statistical Analysis 22: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-0.7 to 16.9] — [estimate comment as in outcome 10, analysis 20]
Statistical Analysis 23: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — CDAI, Week 40. Difference to Placebo for Week 40 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 24: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [0.8 to 20.8] — [estimate comment as in outcome 10, analysis 23]
Statistical Analysis 25: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-0.7 to 16.9] — [estimate comment as in outcome 10, analysis 23]
Statistical Analysis 26: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — CDAI, Week 44. Difference to Placebo for Week 44 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 27: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [0.8 to 20.8] — [estimate comment as in outcome 10, analysis 26]
Statistical Analysis 28: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [0.8 to 20.8] — [estimate comment as in outcome 10, analysis 26]
Statistical Analysis 29: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — CDAI, Week 48. Difference to Placebo for Week 48 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 30: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [2.5 to 24.5] — [estimate comment as in outcome 10, analysis 29]
Statistical Analysis 31: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — [estimate comment as in outcome 10, analysis 29]
Statistical Analysis 32: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [2.5 to 24.5] — CDAI, Week 52. Difference to Placebo for Week 52 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 33: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 10, analysis 32]
Statistical Analysis 34: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-0.7 to 16.9] — CDAI, Week 62 (follow-up). Difference to Placebo for Week 62 (follow-up) is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 35: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — [estimate comment as in outcome 10, analysis 34]
Statistical Analysis 36: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — CDAI, Week 2. Difference to Placebo for Week 2 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction
Statistical Analysis 37: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — CDAI, Week 4. Difference to Placebo for Week 4 is presented. 95% CI were constructed using asymptotic Wald confidence limits without correction.6
Statistical Analysis 38: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — [estimate comment as in outcome 10, analysis 2]
Statistical Analysis 39: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — [estimate comment as in outcome 10, analysis 2]
Statistical Analysis 40: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 0.0, 95% CI 2-sided [-7.4 to 7.4] — [estimate comment as in outcome 10, analysis 3]
Statistical Analysis 41: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 0.0, 95% CI 2-sided [-7.4 to 7.4] — [estimate comment as in outcome 10, analysis 3]
Statistical Analysis 42: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 0.0, 95% CI 2-sided [-7.4 to 7.4] — [estimate comment as in outcome 10, analysis 6]
Statistical Analysis 43: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-6.3 to 11.7] — [estimate comment as in outcome 10, analysis 6]
Statistical Analysis 44: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — [estimate comment as in outcome 10, analysis 9]
Statistical Analysis 45: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; 5.4 = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 10, analysis 9]
Statistical Analysis 46: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 2.7, 95% CI 2-sided [-2.5 to 7.9] — [estimate comment as in outcome 10, analysis 12]
Statistical Analysis 47: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 10, analysis 12]
Statistical Analysis 48: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-0.7 to 16.9] — [estimate comment as in outcome 10, analysis 14]
Statistical Analysis 49: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 10, analysis 14]
Statistical Analysis 50: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [2.5 to 24.5] — [estimate comment as in outcome 10, analysis 16]
Statistical Analysis 51: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-0.7 to 16.9] — [estimate comment as in outcome 10, analysis 18]
Statistical Analysis 52: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [0.8 to 20.8] — [estimate comment as in outcome 10, analysis 18]
Statistical Analysis 53: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [2.5 to 24.5] — [estimate comment as in outcome 10, analysis 20]
Statistical Analysis 54: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 10, analysis 20]
Statistical Analysis 55: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 10, analysis 23]
Statistical Analysis 56: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 13.5, 95% CI 2-sided [2.5 to 24.5] — [estimate comment as in outcome 10, analysis 23]
Statistical Analysis 57: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 10, analysis 26]
Statistical Analysis 58: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 10, analysis 26]
Statistical Analysis 59: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 10.8, 95% CI 2-sided [0.8 to 20.8] — [estimate comment as in outcome 10, analysis 29]
Statistical Analysis 60: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-0.7 to 16.9] — [estimate comment as in outcome 10, analysis 29]
Statistical Analysis 61: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 10, analysis 32]
Statistical Analysis 62: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 8.1, 95% CI 2-sided [-0.7 to 16.9] — [estimate comment as in outcome 10, analysis 32]
Statistical Analysis 63: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 10, analysis 34]
Statistical Analysis 64: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Difference = 16.2, 95% CI 2-sided [4.3 to 28.1] — [estimate comment as in outcome 10, analysis 34]
Statistical Analysis 65: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; Difference = 5.4, 95% CI 2-sided [-1.9 to 12.7] — [estimate comment as in outcome 6, analysis 28]

11. Secondary Outcome: Change From Baseline in SDAI at All Assessment Time Points
Description: SDAI combines information relating to the number of swollen and tender joints, in addition to a measure of general health from both the participants and the physician and acute phase reactants. The SDAI utilizing joint scores from the following 28 joints: elbows, shoulders, elbow, wrists, metacarpal-phalangeal I-V, proximal interphalangeal I-V and knees. It is calculated using the following formula: SDAI = TJC28 + SJC28 + GH + GP + CRP Where TJC - Tender joint Count, SJC= Swollen Joint Count, (GH=participant assessment, GP= physician assessment of disease activity using a 10 centimetre [cm] visual analogue scale [VAS] with 0 = best, 10 = worst), and CRP= C reactive Protein (in mg/L). It ranges between 0.1 and 86. High score indicates worse outcome, low score indicates better outcome. Baseline was defined as the last available assessment prior to the start of study treatment. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline and Weeks 1, 2, 4, 6, 8, 12, 16, 20 and 24
Population: ITT Population. Only those participants available at the specified time points were analyzed (represented by n=x in the category titles).
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | GSK3196165 22.5 mg | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 135 mg | GSK3196165 180 mg
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37 | 37
Scores on a scale
  SDAI, Week 1,n=35,36,32,35, 34, 37: number analyzed (Participants) | 35 | 36 | 32 | 35 | 34 | 37
  SDAI, Week 1,n=35,36,32,35, 34, 37 | -1.53 (1.470) | -5.62 (1.466) | -5.20 (1.527) | -5.86 (1.470) | -6.31 (1.495) | -9.30 (1.448)
  SDAI, Week 2,n=35,34,34,36,36,36: number analyzed (Participants) | 35 | 34 | 34 | 36 | 36 | 36
  SDAI, Week 2,n=35,34,34,36,36,36 | -4.56 (1.821) | -8.62 (1.848) | -9.28 (1.851) | -10.03 (1.804) | -11.22 (1.819) | -11.40 (1.808)
  SDAI, Week 4,n=32,33,34,35, 36, 36: number analyzed (Participants) | 32 | 33 | 34 | 35 | 36 | 36
  SDAI, Week 4,n=32,33,34,35, 36, 36 | -5.53 (2.095) | -12.30 (2.092) | -12.81 (2.073) | -14.76 (2.037) | -13.97 (2.042) | -18.03 (2.032)
  SDAI, Week 6,n=35,34,33,36,32, 36: number analyzed (Participants) | 35 | 34 | 33 | 36 | 32 | 36
  SDAI, Week 6,n=35,34,33,36,32, 36 | -8.70 (2.132) | -14.36 (2.152) | -14.99 (2.163) | -15.50 (2.095) | -15.70 (2.165) | -18.86 (2.109)
  SDAI, Week 8,n=34,33,34,37, 35, 32: number analyzed (Participants) | 34 | 33 | 34 | 37 | 35 | 32
  SDAI, Week 8,n=34,33,34,37, 35, 32 | -8.08 (2.349) | -14.66 (2.367) | -17.23 (2.353) | -16.95 (2.281) | -19.26 (2.329) | -22.09 (2.358)
  SDAI, Week 12,n=34,35,33,37, 34, 36: number analyzed (Participants) | 34 | 35 | 33 | 37 | 34 | 36
  SDAI, Week 12,n=34,35,33,37, 34, 36 | -7.05 (2.729) | -13.95 (2.712) | -17.41 (2.741) | -21.20 (2.640) | -16.73 (2.708) | -23.90 (2.676)
  SDAI, Week 16,n=8,16,20,23, 18, 36: number analyzed (Participants) | 8 | 16 | 20 | 23 | 18 | 36
  SDAI, Week 16,n=8,16,20,23, 18, 36 | -15.64 (3.222) | -17.53 (2.707) | -22.64 (2.605) | -22.91 (2.484) | -21.68 (2.632) | -25.08 (2.351)
  SDAI, Week 20,n=8,15,20,25, 18, 35: number analyzed (Participants) | 8 | 15 | 20 | 25 | 18 | 35
  SDAI, Week 20,n=8,15,20,25, 18, 35 | -17.47 (3.523) | -16.67 (2.835) | -23.17 (2.621) | -23.47 (2.437) | -24.06 (2.670) | -26.17 (2.263)
  SDAI, Week 24,n=8,14,20,24, 19, 33: number analyzed (Participants) | 8 | 14 | 20 | 24 | 19 | 33
  SDAI, Week 24,n=8,14,20,24, 19, 33 | -5.40 (4.484) | -16.05 (3.569) | -21.77 (3.165) | -21.07 (2.945) | -21.28 (3.200) | -26.27 (2.667)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.050, MMRM — MMRM analysis adjusted for SDAI Baseline score, treatment group, visit and treatment group by visit and Baseline by visit interactions; Mean Difference (Net) = -4.09, 95% CI 2-sided [-8.18 to 0.00] — Week 1, SDAI
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.086, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -3.66, 95% CI 2-sided [-7.84 to 0.52] — Week 1,SDAI
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.038, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -4.33, 95% CI 2-sided [-8.43 to -0.23] — Week 1,SDAI
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.119, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -4.06, 95% CI 2-sided [-9.18 to 1.05] — Week 2,SDAI
Statistical Analysis 5: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.071, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -4.72, 95% CI 2-sided [-9.85 to 0.40] — Week 2,SDAI
Statistical Analysis 6: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.034, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -5.48, 95% CI 2-sided [-10.53 to -0.42] — Week 2,SDAI
Statistical Analysis 7: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.023, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -6.78, 95% CI 2-sided [-12.61 to -0.94] — Week 4,SDAI
Statistical Analysis 8: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.014, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -7.28, 95% CI 2-sided [-13.09 to -1.47] — Week 4,SDAI
Statistical Analysis 9: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.002, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -9.23, 95% CI 2-sided [-14.99 to -3.47] — Week 4,SDAI
Statistical Analysis 10: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.063, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -5.65, 95% CI 2-sided [-11.62 to 0.32] — Week 6,SDAI
Statistical Analysis 11: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.040, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -6.29, 95% CI 2-sided [-12.28 to -0.30] — Week 6,SDAI
Statistical Analysis 12: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.024, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -6.79, 95% CI 2-sided [-12.69 to -0.90] — Week 6,SDAI
Statistical Analysis 13: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.050, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -6.58, 95% CI 2-sided [-13.15 to -0.01] — Week 8,SDAI
Statistical Analysis 14: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.006, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -9.15, 95% CI 2-sided [-15.71 to -2.60] — Week 8,SDAI
Statistical Analysis 15: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.007, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -8.86, 95% CI 2-sided [-15.32 to -2.41] — Week 8,SDAI
Statistical Analysis 16: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.074, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -6.91, 95% CI 2-sided [-14.49 to 0.68] — Week 12,SDAI
Statistical Analysis 17: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.008, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -10.37, 95% CI 2-sided [-17.99 to -2.74] — Week 12,SDAI
Statistical Analysis 18: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p < 0.001, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -14.15, 95% CI 2-sided [-21.64 to -6.67] — Week 12,SDAI
Statistical Analysis 19: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.656, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -1.88, 95% CI 2-sided [-10.19 to 6.43] — Week 16,SDAI
Statistical Analysis 20: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.093, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -7.00, 95% CI 2-sided [-15.19 to 1.19] — Week 16,SDAI
Statistical Analysis 21: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.076, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -7.26, 95% CI 2-sided [-15.30 to 0.78] — Week 16,SDAI
Statistical Analysis 22: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.860, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = 0.80, 95% CI 2-sided [-8.14 to 9.74] — Week 20,SDAI
Statistical Analysis 23: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.196, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -5.71, 95% CI 2-sided [-14.40 to 2.99] — Week 20,SDAI
Statistical Analysis 24: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.164, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -6.00, 95% CI 2-sided [-14.48 to 2.48] — Week 20,SDAI
Statistical Analysis 25: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.066, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -10.65, 95% CI 2-sided [-21.99 to 0.69] — Week 24,SDAI
Statistical Analysis 26: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.003, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -16.37, 95% CI 2-sided [-27.25 to -5.49] — Week 24,SDAI
Statistical Analysis 27: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.004, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -15.67, 95% CI 2-sided [-26.30 to -5.03] — Week 24,SDAI
Statistical Analysis 28: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.024, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -4.78, 95% CI 2-sided [-8.91 to -0.65] — Week 1,SDAI
Statistical Analysis 29: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p < 0.001, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -7.77, 95% CI 2-sided [-11.84 to -3.70] — Week 1,SDAI
Statistical Analysis 30: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.010, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -6.67, 95% CI 2-sided [-11.74 to -1.60] — Week 2,SDAI
Statistical Analysis 31: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.008, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -6.85, 95% CI 2-sided [-11.91 to -1.78] — Week 2,SDAI
Statistical Analysis 32: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.004, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -8.44, 95% CI 2-sided [-14.20 to -2.67] — Week 4,SDAI
Statistical Analysis 33: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p < 0.001, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -12.51, 95% CI 2-sided [-18.26 to -6.75] — Week 4,SDAI
Statistical Analysis 34: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.022, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -7.00, 95% CI 2-sided [-12.99 to -1.01] — Week 6,SDAI
Statistical Analysis 35: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p < 0.001, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -10.16, 95% CI 2-sided [-16.07 to -4.24] — Week 6,SDAI
Statistical Analysis 36: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p < 0.001, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -11.18, 95% CI 2-sided [-17.70 to -4.66] — Week 8,SDAI
Statistical Analysis 37: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p < 0.001, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -14.00, 95% CI 2-sided [-20.57 to -7.44] — Week 8,SDAI
Statistical Analysis 38: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.013, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -9.68, 95% CI 2-sided [-17.26 to -2.11] — Week 12,SDAI
Statistical Analysis 39: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p < 0.001, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -16.86, 95% CI 2-sided [-24.39 to -9.32] — Week 12,SDAI
Statistical Analysis 40: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.149, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -6.03, 95% CI 2-sided [-14.24 to 2.18] — Week 16,SDAI
Statistical Analysis 41: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.019, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -9.43, 95% CI 2-sided [-17.32 to -1.55] — Week 16,SDAI
Statistical Analysis 42: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.138, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -6.59, 95% CI 2-sided [-15.32 to 2.14] — Week 20,SDAI
Statistical Analysis 43: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.040, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -8.70, 95% CI 2-sided [-16.99 to -0.42] — Week 20,SDAI
Statistical Analysis 44: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.005, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -15.88, 95% CI 2-sided [-26.77 to -4.98] — Week 24,SDAI
Statistical Analysis 45: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p < 0.001, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -20.87, 95% CI 2-sided [-31.20 to -10.53] — Week 24,SDAI

12. Secondary Outcome: Change From Baseline in CDAI at All Assessment Time Points
Description: CDAI combines information relating to the number of swollen and tender joints, in addition to a measure of general health from both the participants and the physician. CDAI utilizing joint scores from the following 28 joints: elbows, shoulders, elbow, wrists, metacarpal- phalangeal I-V, proximal interphalangeal I-V and knees and is calculated using the following formula: CDAI =TJC28 + SJC28 + GH + GP Where TJC - Tender joint Count, SJC= Swollen Joint Count, (GH=participant assessment of disease activity and GP=physician assessment of disease activity using a 10 cm visual analogue scale with 0 = best, 100 = worst). It ranges between 0 and 76. High score indicates worse outcome, low score indicates better outcome. Baseline was defined as the last available assessment prior to the start of study treatment. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline and Weeks 1, 2, 4, 6, 8, 12, 16, 20 and 24
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | GSK3196165 22.5 mg | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 135 mg | GSK3196165 180 mg
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37 | 37
Scores on a scale
  CDAI, Week 1, n=36,36,33,36, 35, 37: number analyzed (Participants) | 36 | 36 | 33 | 36 | 35 | 37
  CDAI, Week 1, n=36,36,33,36, 35, 37 | -1.34 (1.449) | -5.18 (1.455) | -5.18 (1.497) | -5.76 (1.448) | -5.23 (1.469) | -8.73 (1.438)
  CDAI, Week 2,n=35,34,36,37, 36, 37: number analyzed (Participants) | 35 | 34 | 36 | 37 | 36 | 37
  CDAI, Week 2,n=35,34,36,37, 36, 37 | -4.25 (1.782) | -8.42 (1.807) | -7.72 (1.771) | -9.45 (1.752) | -10.35 (1.777) | -11.10 (1.755)
  CDAI, Week 4,n=33,33,35,36, 36, 36: number analyzed (Participants) | 33 | 33 | 35 | 36 | 36 | 36
  CDAI, Week 4,n=33,33,35,36, 36, 36 | -4.95 (2.013) | -12.15 (2.024) | -11.68 (1.978) | -14.15 (1.958) | -12.88 (1.974) | -17.14 (1.965)
  CDAI, Week 6,n=35,35,33,37, 34, 36: number analyzed (Participants) | 35 | 35 | 33 | 37 | 34 | 36
  CDAI, Week 6,n=35,35,33,37, 34, 36 | -8.20 (2.089) | -13.68 (2.094) | -14.05 (2.101) | -14.83 (2.042) | -13.82 (2.094) | -18.37 (2.065)
  CDAI, Week 8,n=34,33,35,37, 35, 34: number analyzed (Participants) | 34 | 33 | 35 | 37 | 35 | 34
  CDAI, Week 8,n=34,33,35,37, 35, 34 | -7.57 (2.298) | -13.98 (2.315) | -16.17 (2.270) | -16.31 (2.232) | -17.94 (2.276) | -21.36 (2.279)
  CDAI, Week 12,n=34,35,35,37, 35, 36: number analyzed (Participants) | 34 | 35 | 35 | 37 | 35 | 36
  CDAI, Week 12,n=34,35,35,37, 35, 36 | -6.59 (2.658) | -13.40 (2.640) | -16.39 (2.621) | -20.47 (2.571) | -16.26 (2.625) | -23.23 (2.604)
  CDAI, Week 16,n=8,16,21,23, 18, 36: number analyzed (Participants) | 8 | 16 | 21 | 23 | 18 | 36
  CDAI, Week 16,n=8,16,21,23, 18, 36 | -15.61 (3.077) | -17.30 (2.586) | -21.94 (2.445) | -22.05 (2.371) | -21.14 (2.508) | -24.47 (2.245)
  CDAI, Week 20,n=8,15,21,25, 18, 35: number analyzed (Participants) | 8 | 15 | 21 | 25 | 18 | 35
  CDAI, Week 20,n=8,15,21,25, 18, 35 | -16.91 (3.419) | -15.87 (2.730) | -22.31 (2.470) | -22.81 (2.334) | -23.46 (2.564) | -25.58 (2.158)
  CDAI, Week 24,n=8,14,21,24, 19, 33: number analyzed (Participants) | 8 | 14 | 21 | 24 | 19 | 33
  CDAI, Week 24,n=8,14,21,24, 19, 33 | -5.77 (4.267) | -15.14 (3.389) | -20.88 (2.947) | -20.67 (2.791) | -21.19 (3.037) | -25.65 (2.529)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.063, MMRM — MMRM analysis adjusted for CDAI Baseline score, treatment group, visit and treatment group by visit and Baseline by visit interactions; Mean Difference (Net) = -3.84, 95% CI 2-sided [-7.89 to 0.20] — Week 1,CDAI
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.067, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -3.84, 95% CI 2-sided [-7.95 to 0.28] — Week 1,CDAI
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.032, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -4.43, 95% CI 2-sided [-8.46 to -0.39] — Week 1,CDAI
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.102, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -4.17, 95% CI 2-sided [-9.17 to 0.84] — Week 2,CDAI
Statistical Analysis 5: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.170, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -3.47, 95% CI 2-sided [-8.43 to 1.49] — Week 2,CDAI
Statistical Analysis 6: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.039, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -5.20, 95% CI 2-sided [-10.13 to -0.27] — Week 2,CDAI
Statistical Analysis 7: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.012, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -7.20, 95% CI 2-sided [-12.82 to -1.57] — Week 4,CDAI
Statistical Analysis 8: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.018, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -6.73, 95% CI 2-sided [-12.30 to -1.16] — Week 4,CDAI
Statistical Analysis 9: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.001, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -9.19, 95% CI 2-sided [-14.73 to -3.66] — Week 4,CDAI
Statistical Analysis 10: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.065, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -5.48, 95% CI 2-sided [-11.31 to 0.35] — Week 6,CDAI
Statistical Analysis 11: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.050, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -5.85, 95% CI 2-sided [-11.69 to -0.00] — Week 6,CDAI
Statistical Analysis 12: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.024, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Final Values) = -6.63, 95% CI 2-sided [-12.38 to -0.87] — Week 6,CDAI
Statistical Analysis 13: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.051, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -6.41, 95% CI 2-sided [-12.84 to 0.02] — Week 8,CDAI
Statistical Analysis 14: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.008, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -8.60, 95% CI 2-sided [-14.97 to -2.22] — Week 8,CDAI
Statistical Analysis 15: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.007, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -8.74, 95% CI 2-sided [-15.06 to -2.43] — Week 8,CDAI
Statistical Analysis 16: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.071, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -6.80, 95% CI 2-sided [-14.19 to 0.58] — Week 12,CDAI
Statistical Analysis 17: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.009, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -9.80, 95% CI 2-sided [-17.17 to -2.44] — Week 12,CDAI
Statistical Analysis 18: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p < 0.001, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -13.88, 95% CI 2-sided [-21.17 to -6.59] — Week 12,CDAI
Statistical Analysis 19: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.676, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -1.68, 95% CI 2-sided [-9.63 to 6.26] — Week 16,CDAI
Statistical Analysis 20: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.110, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -6.33, 95% CI 2-sided [-14.11 to 1.44] — Week 16,CDAI
Statistical Analysis 21: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.099, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -6.44, 95% CI 2-sided [-14.12 to 1.23] — Week 16,CDAI
Statistical Analysis 22: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.812, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = 1.04, 95% CI 2-sided [-7.61 to 9.69] — Week 20,CDAI
Statistical Analysis 23: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.204, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -5.39, 95% CI 2-sided [-13.75 to 2.96] — Week 20,CDAI
Statistical Analysis 24: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.157, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -5.90, 95% CI 2-sided [-14.09 to 2.30] — Week 20,CDAI
Statistical Analysis 25: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.088, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -9.37, 95% CI 2-sided [-20.15 to 1.42] — Week 24,CDAI
Statistical Analysis 26: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.004, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -15.12, 95% CI 2-sided [-25.40 to -4.83] — Week 24,CDAI
Statistical Analysis 27: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.004, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -14.91, 95% CI 2-sided [-25.01 to -4.80] — Week 24,CDAI
Statistical Analysis 28: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.060, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -3.89, 95% CI 2-sided [-7.96 to 0.17] — Week 1,CDAI
Statistical Analysis 29: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p < 0.001, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -7.39, 95% CI 2-sided [-11.42 to -3.36] — Week 1,CDAI
Statistical Analysis 30: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.016, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -6.10, 95% CI 2-sided [-11.06 to -1.14] — Week 2,CDAI
Statistical Analysis 31: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.007, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -6.85, 95% CI 2-sided [-11.78 to -1.91] — Week 2,CDAI
Statistical Analysis 32: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.005, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -7.92, 95% CI 2-sided [-13.48 to -2.37] — Week 4,CDAI
Statistical Analysis 33: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p < 0.001, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -12.19, 95% CI 2-sided [-17.74 to -6.64] — Week 4,CDAI
Statistical Analysis 34: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.059, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -5.62, 95% CI 2-sided [-11.45 to 0.21] — Week 6,CDAI
Statistical Analysis 35: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p < 0.001, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -10.17, 95% CI 2-sided [-15.97 to -4.38] — Week 6,CDAI
Statistical Analysis 36: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.002, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -10.37, 95% CI 2-sided [-16.75 to -4.00] — Week 8,CDAI
Statistical Analysis 37: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p < 0.001, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -13.79, 95% CI 2-sided [-20.18 to -7.41] — Week 8,CDAI
Statistical Analysis 38: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.010, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -9.67, 95% CI 2-sided [-17.03 to -2.31] — Week 12,CDAI
Statistical Analysis 39: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p < 0.001, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -16.63, 95% CI 2-sided [-23.97 to -9.30] — Week 12,CDAI
Statistical Analysis 40: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.165, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -5.53, 95% CI 2-sided [-13.37 to 2.30] — Week 16,CDAI
Statistical Analysis 41: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.022, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -8.85, 95% CI 2-sided [-16.39 to -1.32] — Week 16,CDAI
Statistical Analysis 42: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.127, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -6.55, 95% CI 2-sided [-14.99 to 1.89] — Week 20,CDAI
Statistical Analysis 43: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.034, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -8.67, 95% CI 2-sided [-16.67 to -0.67] — Week 20,CDAI
Statistical Analysis 44: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.004, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -15.43, 95% CI 2-sided [-25.78 to -5.07] — Week 24,CDAI
Statistical Analysis 45: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p < 0.001, MMRM — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -19.88, 95% CI 2-sided [-29.70 to -10.06] — Week 24,CDAI

13. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) at All Assessment Time Points
Description: HAQ-DI is 20-question instrument that assesses the degree of difficulty a person has in accomplishing tasks in eight functional areas;dressing and grooming, arising, eating, walking, hygiene, reach, grip, and common daily activities. Each functional area contains at least two questions. For each question, there is a four level response set that is scored from 0 (without any difficulty) to 3 (unable to do). If aids or devices or physical assistance are used for a specific functional area and the maximum response of this functional area is 0 or 1 the according value is increased to a score of 2. HAQ-DI is only calculated if there are at least 6 functional area scores available. The average of these non-missing functional area scores defines the continuous HAQ-DI score ranging from 0 to 3. Baseline was defined as the last available assessment prior to the start of study treatment. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline and Weeks 1, 2, 4, 6, 8, 12, 16, 20 and 24
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | GSK3196165 22.5 mg | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 135 mg | GSK3196165 180 mg
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37 | 37
Scores on a scale
  HAQ-DI, Week 1,n=36,36,35,36, 36, 37: number analyzed (Participants) | 36 | 36 | 35 | 36 | 36 | 37
  HAQ-DI, Week 1,n=36,36,35,36, 36, 37 | -0.09 (0.054) | -0.08 (0.054) | -0.08 (0.054) | -0.10 (0.054) | -0.13 (0.054) | -0.17 (0.053)
  HAQ-DI, Week 2,n=36,35,37,37, 36, 37: number analyzed (Participants) | 36 | 35 | 37 | 37 | 36 | 37
  HAQ-DI, Week 2,n=36,35,37,37, 36, 37 | -0.17 (0.062) | -0.13 (0.063) | -0.16 (0.062) | -0.23 (0.062) | -0.25 (0.063) | -0.26 (0.062)
  HAQ-DI, Week 4,n=34,34,36,37, 36, 36: number analyzed (Participants) | 34 | 34 | 36 | 37 | 36 | 36
  HAQ-DI, Week 4,n=34,34,36,37, 36, 36 | -0.22 (0.073) | -0.18 (0.073) | -0.17 (0.072) | -0.29 (0.071) | -0.29 (0.072) | -0.40 (0.072)
  HAQ-DI, Week 6,n=35,35,35,37, 36, 36: number analyzed (Participants) | 35 | 35 | 35 | 37 | 36 | 36
  HAQ-DI, Week 6,n=35,35,35,37, 36, 36 | -0.23 (0.077) | -0.22 (0.077) | -0.27 (0.077) | -0.33 (0.076) | -0.21 (0.077) | -0.43 (0.076)
  HAQ-DI, Week 8,n=34,34,35,37, 35, 34: number analyzed (Participants) | 34 | 34 | 35 | 37 | 35 | 34
  HAQ-DI, Week 8,n=34,34,35,37, 35, 34 | -0.22 (0.082) | -0.18 (0.082) | -0.33 (0.081) | -0.31 (0.080) | -0.35 (0.081) | -0.42 (0.081)
  HAQ-DI, Week 12,n=34,35, 35, 37,35, 36: number analyzed (Participants) | 34 | 35 | 35 | 37 | 35 | 36
  HAQ-DI, Week 12,n=34,35, 35, 37,35, 36 | -0.26 (0.091) | -0.31 (0.091) | -0.30 (0.090) | -0.37 (0.89) | -0.38 (0.090) | -0.50 (0.090)
  HAQ-DI, Week 16,n=8,16,21,24, 18, 36: number analyzed (Participants) | 8 | 16 | 21 | 24 | 18 | 36
  HAQ-DI, Week 16,n=8,16,21,24, 18, 36 | -0.49 (0.141) | -0.33 (0.111) | -0.38 (0.102) | -0.57 (0.098) | -0.40 (0.106) | -0.50 (0.090)
  HAQ-DI, Week 20,n=8,15,21,25, 19, 36: number analyzed (Participants) | 8 | 15 | 21 | 25 | 19 | 36
  HAQ-DI, Week 20,n=8,15,21,25, 19, 36 | -0.35 (0.139) | -0.37 (0.112) | -0.42 (0.103) | -0.51 (0.097) | -0.49 (0.105) | -0.56 (0.091)
  HAQ-DI, Week 24,n=8,14,21,24, 19, 34: number analyzed (Participants) | 8 | 14 | 21 | 24 | 19 | 34
  HAQ-DI, Week 24,n=8,14,21,24, 19, 34 | -0.34 (0.143) | -0.32 (0.116) | -0.41 (0.104) | -0.43 (0.099) | -0.42 (0.107) | -0.54 (0.092)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.938, MMRM — MMRM analysis adjusted for HAQ-DI Baseline score, treatment group, visit and treatment group by visit and Baseline by visit interactions; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.14 to 0.16] — Week 1, HAQ-DI
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.981, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = 0.00, 95% CI 2-sided [-0.15 to 0.15] — Week 1, HAQ-DI
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.857, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.16 to 0.14] — Week 1, HAQ-DI
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.592, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = 0.05, 95% CI 2-sided [-0.13 to 0.22] — Week 2, HAQ-DI
Statistical Analysis 5: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.917, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.16 to 0.18] — Week 2, HAQ-DI
Statistical Analysis 6: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.545, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = -0.05, 95% CI 2-sided [-0.23 to 0.12] — Week 2, HAQ-DI
Statistical Analysis 7: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.707, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = 0.04, 95% CI 2-sided [-0.16 to 0.24] — Week 4, HAQ-DI
Statistical Analysis 8: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.603, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = 0.05, 95% CI 2-sided [-0.15 to 0.26] — Week 4, HAQ-DI
Statistical Analysis 9: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.473, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.27 to 0.13] — Week 4, HAQ-DI
Statistical Analysis 10: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.987, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = 0.00, 95% CI 2-sided [-0.21 to 0.22] — Week 6, HAQ-DI
Statistical Analysis 11: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.713, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = -0.04, 95% CI 2-sided [-0.25 to 0.17] — Week 6, HAQ-DI
Statistical Analysis 12: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.357, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = -0.10, 95% CI 2-sided [-0.31 to 0.11] — Week 6, HAQ-DI
Statistical Analysis 13: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.748, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.19 to 0.26] — Week 8, HAQ-DI
Statistical Analysis 14: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.327, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = -0.11, 95% CI 2-sided [-0.34 to 0.11] — Week 8, HAQ-DI
Statistical Analysis 15: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.395, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = -0.10, 95% CI 2-sided [-0.32 to 0.13] — Week 8, HAQ-DI
Statistical Analysis 16: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.710, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = -0.05, 95% CI 2-sided [-0.30 to 0.21] — Week 12, HAQ-DI
Statistical Analysis 17: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.740, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = -0.04, 95% CI 2-sided [-0.30 to 0.21] — Week 12, HAQ-DI
Statistical Analysis 18: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.398, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = -0.11, 95% CI 2-sided [-0.36 to 0.14] — Week 12, HAQ-DI
Statistical Analysis 19: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.364, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = 0.16, 95% CI 2-sided [-0.19 to 0.52] — Week 16, HAQ-DI
Statistical Analysis 20: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.503, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = 0.12, 95% CI 2-sided [-0.23 to 0.46] — Week 16, HAQ-DI
Statistical Analysis 21: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.647, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = -0.08, 95% CI 2-sided [-0.42 to 0.26] — Week 16, HAQ-DI
Statistical Analysis 22: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.910, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.37 to 0.33] — Week 20, HAQ-DI
Statistical Analysis 23: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.660, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = -0.08, 95% CI 2-sided [-0.42 to 0.26] — Week 20, HAQ-DI
Statistical Analysis 24: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.340, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = -0.16, 95% CI 2-sided [-0.50 to 0.17] — Week 20, HAQ-DI
Statistical Analysis 25: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.902, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = 0.02, 95% CI 2-sided [-0.34 to 0.39] — Week 24, HAQ-DI
Statistical Analysis 26: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.687, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.42 to 0.28] — Week 24, HAQ-DI
Statistical Analysis 27: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.599, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = -0.09, 95% CI 2-sided [-0.44 to 0.25] — Week 24, HAQ-DI
Statistical Analysis 28: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.588, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = -0.04, 95% CI 2-sided [-0.19 to 0.11] — Week 1, HAQ-DI
Statistical Analysis 29: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.259, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = -0.09, 95% CI 2-sided [-0.23 to 0.06] — Week 1, HAQ-DI
Statistical Analysis 30: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.358, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = -0.08, 95% CI 2-sided [-0.26 to 0.09] — Week 2, HAQ-DI
Statistical Analysis 31: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.325, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = -0.09, 95% CI 2-sided [-0.26 to 0.09] — Week 2, HAQ-DI
Statistical Analysis 32: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.473, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.28 to 0.13] — Week 4, HAQ-DI
Statistical Analysis 33: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.085, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = -0.18, 95% CI 2-sided [-0.38 to 0.02] — Week 4, HAQ-DI
Statistical Analysis 34: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.897, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.20 to 0.23] — Week 6, HAQ-DI
Statistical Analysis 35: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.065, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = -0.20, 95% CI 2-sided [-0.42 to 0.01] — Week 6, HAQ-DI
Statistical Analysis 36: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.238, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = -0.14, 95% CI 2-sided [-0.36 to 0.09] — Week 8, HAQ-DI
Statistical Analysis 37: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.071, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = -0.21, 95% CI 2-sided [-0.44 to 0.02] — Week 8, HAQ-DI
Statistical Analysis 38: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.340, MMRM — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -0.12, 95% CI 2-sided [-0.38 to 0.13] — Week 12, HAQ-DI
Statistical Analysis 39: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.059, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = -0.24, 95% CI 2-sided [-0.49 to 0.01] — Week 12, HAQ-DI
Statistical Analysis 40: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.607, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = 0.09, 95% CI 2-sided [-0.26 to 0.44] — Week 16, HAQ-DI
Statistical Analysis 41: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.959, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.34 to 0.32] — Week 16, HAQ-DI
Statistical Analysis 42: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.401, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = -0.15, 95% CI 2-sided [-0.49 to 0.20] — Week 20, HAQ-DI
Statistical Analysis 43: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.207, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = -0.21, 95% CI 2-sided [-0.54 to 0.12] — Week 20, HAQ-DI
Statistical Analysis 44: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.637, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Net) = -0.08, 95% CI 2-sided [-0.44 to 0.27] — Week 24, HAQ-DI
Statistical Analysis 45: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.251, MMRM — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.53 to 0.14] — Week 24, HAQ-DI

14. Secondary Outcome: Change From Baseline in Pain Score at All Assessment Time Points
Description: Participants assessed the severity of their current arthritis pain using a 100 unit visual analog scale (VAS) by placing a mark on the scale between 0 (no pain) and 100 (most severe pain), which corresponds to the magnitude of their pain. Baseline was defined as the last available assessment prior to the start of study treatment. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline and Weeks 1, 2, 4, 6, 8, 12, 16, 20 and Week 24
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | GSK3196165 22.5 mg | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 135 mg | GSK3196165 180 mg
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37 | 37
Scores on a scale
  Week 1,n=36,36,35,36, 36,37: number analyzed (Participants) | 36 | 36 | 35 | 36 | 36 | 37
  Week 1,n=36,36,35,36, 36,37 | -2.25 (2.625) | -4.71 (2.648) | -5.02 (2.656) | -9.96 (2.626) | -7.18 (2.637) | -7.89 (2.619)
  Week 2,n=36,35,37,37,36,37: number analyzed (Participants) | 36 | 35 | 37 | 37 | 36 | 37
  Week 2,n=36,35,37,37,36,37 | -3.79 (2.818) | -6.71 (2.870) | -9.77 (2.797) | -11.37 (2.791) | -11.63 (2.829) | -14.22 (2.810)
  Week 4,n=34,34,36,37, 36,36: number analyzed (Participants) | 34 | 34 | 36 | 37 | 36 | 36
  Week 4,n=34,34,36,37, 36,36 | -5.44 (3.081) | -8.47 (3.107) | -14.83 (3.029) | -17.65 (2.995) | -13.39 (3.036) | -19.40 (3.038)
  Week 6,n=35,35,35,37, 36, 36: number analyzed (Participants) | 35 | 35 | 35 | 37 | 36 | 36
  Week 6,n=35,35,35,37, 36, 36 | -6.69 (3.334) | -11.18 (3.357) | -14.71 (3.319) | -15.05 (3.262) | -14.05 (3.306) | -19.12 (3.311)
  Week 8,n=34,34,35,37, 35,34: number analyzed (Participants) | 34 | 34 | 35 | 37 | 35 | 34
  Week 8,n=34,34,35,37, 35,34 | -3.98 (3.555) | -9.60 (3.577) | -18.55 (3.517) | -17.92 (3.461) | -20.49 (3.523) | -24.38 (3.541)
  Week 12,n=34, 35,35,37, 35, 36: number analyzed (Participants) | 34 | 35 | 35 | 37 | 35 | 36
  Week 12,n=34, 35,35,37, 35, 36 | -7.07 (3.705) | -14.09 (3.702) | -21.22 (3.659) | -25.25 (3.593) | -19.07 (3.662) | -25.01 (3.650)
  Week 16,n=8,16,21,24, 18, 16: number analyzed (Participants) | 8 | 16 | 21 | 24 | 18 | 16
  Week 16,n=8,16,21,24, 18, 16 | -12.60 (6.077) | -17.50 (4.768) | -28.56 (4.361) | -26.46 (4.187) | -25.80 (4.549) | -24.48 (3.807)
  Week 20,n=8,15,21,25, 19,36: number analyzed (Participants) | 8 | 15 | 21 | 25 | 19 | 36
  Week 20,n=8,15,21,25, 19,36 | -13.95 (5.589) | -14.64 (4.495) | -27.12 (4.068) | -27.44 (3.870) | -27.86 (4.179) | -27.17 (3.584)
  Week 24,n=8,14,21,24, 19, 34: number analyzed (Participants) | 8 | 14 | 21 | 24 | 19 | 34
  Week 24,n=8,14,21,24, 19, 34 | -13.38 (6.484) | -19.76 (5.231) | -23.52 (4.620) | -25.45 (4.409) | -26.61 (4.756) | -30.08 (4.048)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.511, MMRM — MMRM analysis adjusted for Pain Baseline score, treatment group, visit and treatment group by visit and Baseline by visit interactions; Mean Difference (Net) = -2.45, 95% CI 2-sided [-9.81 to 4.90] — Week 1, Pain score
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.461, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -2.76, 95% CI 2-sided [-10.13 to 4.60] — Week 1, Pain score
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.039, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -7.71, 95% CI 2-sided [-15.03 to -0.39] — Week 1, Pain score
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.469, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -2.92, 95% CI 2-sided [-10.86 to 5.01] — Week 2, Pain score
Statistical Analysis 5: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.133, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -5.99, 95% CI 2-sided [-13.82 to 1.85] — Week 2, Pain score
Statistical Analysis 6: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.057, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -7.58, 95% CI 2-sided [-15.40 to 0.23] — Week 2, Pain score
Statistical Analysis 7: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.490, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -3.03, 95% CI 2-sided [-11.67 to 5.61] — Week 4, Pain score
Statistical Analysis 8: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.031, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -9.38, 95% CI 2-sided [-17.91 to -0.86] — Week 4, Pain score
Statistical Analysis 9: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.005, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -12.21, 95% CI 2-sided [-20.67 to -3.74] — Week 4, Pain score
Statistical Analysis 10: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.345, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -4.49, 95% CI 2-sided [-13.83 to 4.85] — Week 6, Pain score
Statistical Analysis 11: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.090, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -8.02, 95% CI 2-sided [-17.30 to 1.26] — Week 6, Pain score
Statistical Analysis 12: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.074, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -8.36, 95% CI 2-sided [-17.55 to 0.83] — Week 6, Pain score
Statistical Analysis 13: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.268, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -5.61, 95% CI 2-sided [-15.57 to 4.34] — Week 8, Pain score
Statistical Analysis 14: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.004, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -14.57, 95% CI 2-sided [-24.43 to -4.70] — Week 8, Pain score
Statistical Analysis 15: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.005, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -13.94, 95% CI 2-sided [-23.72 to -4.16] — Week 8, Pain score
Statistical Analysis 16: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.182, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -7.02, 95% CI 2-sided [-17.36 to 3.32] — Week 12, Pain score
Statistical Analysis 17: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.007, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -14.15, 95% CI 2-sided [-24.42 to -3.87] — Week 12, Pain score
Statistical Analysis 18: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p < 0.001, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -18.18, 95% CI 2-sided [-28.35 to -8.01] — Week 12, Pain score
Statistical Analysis 19: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.527, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -4.89, 95% CI 2-sided [-20.15 to 10.36] — Week 16, Pain score
Statistical Analysis 20: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.034, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -15.95, 95% CI 2-sided [-30.72 to -1.19] — Week 16, Pain score
Statistical Analysis 21: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.062, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -13.86, 95% CI 2-sided [-28.42 to 0.70] — Week 16, Pain score
Statistical Analysis 22: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.924, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -0.69, 95% CI 2-sided [-14.85 to 13.47] — Week 20, Pain score
Statistical Analysis 23: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.058, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -13.17, 95% CI 2-sided [-26.82 to 0.48] — Week 20, Pain score
Statistical Analysis 24: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.049, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -13.49, 95% CI 2-sided [-26.91 to -0.08] — Week 20, Pain score
Statistical Analysis 25: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.445, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -6.38, 95% CI 2-sided [-22.84 to 10.07] — Week 24, Pain score
Statistical Analysis 26: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.205, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -10.14, 95% CI 2-sided [-25.87 to 5.58] — Week 24, Pain score
Statistical Analysis 27: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.125, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -12.07, 95% CI 2-sided [-27.55 to 3.41] — Week 24, Pain score
Statistical Analysis 28: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.187, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -4.93, 95% CI 2-sided [-12.26 to 2.41] — Week 1, Pain score
Statistical Analysis 29: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.130, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -5.63, 95% CI 2-sided [-12.93 to 1.67] — Week 1, Pain score
Statistical Analysis 30: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.051, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -7.85, 95% CI 2-sided [-15.72 to 0.03] — Week 2, Pain score
Statistical Analysis 31: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.009, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -10.44, 95% CI 2-sided [-18.27 to -2.60] — Week 2, Pain score
Statistical Analysis 32: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.068, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -7.94, 95% CI 2-sided [-16.47 to 0.58] — Week 4, Pain score
Statistical Analysis 33: Comparison: GSK3196165 180 mg; Test type: Other; p = 0.001, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -13.96, 95% CI 2-sided [-22.47 to -5.44] — Week 4, Pain score
Statistical Analysis 34: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.118, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -7.36, 95% CI 2-sided [-16.62 to 1.89] — Week 6, Pain score
Statistical Analysis 35: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.009, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -12.43, 95% CI 2-sided [-21.68 to -3.19] — Week 6, Pain score
Statistical Analysis 36: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.001, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -16.51, 95% CI 2-sided [-26.38 to -6.65] — Week 8, Pain score
Statistical Analysis 37: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p < 0.001, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -20.39, 95% CI 2-sided [-30.27 to -10.52] — Week 8, Pain score
Statistical Analysis 38: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.022, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -12.00, 95% CI 2-sided [-22.27 to -1.73] — Week 12, Pain score
Statistical Analysis 39: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p < 0.001, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -17.94, 95% CI 2-sided [-28.18 to -7.70] — Week 12, Pain score
Statistical Analysis 40: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.084, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -13.20, 95% CI 2-sided [-28.18 to 1.79] — Week 16, Pain score
Statistical Analysis 41: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.099, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -11.87, 95% CI 2-sided [-26.02 to 2.27] — Week 16, Pain score
Statistical Analysis 42: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.048, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -13.91, 95% CI 2-sided [-27.68 to -0.14] — Week 20, Pain score
Statistical Analysis 43: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.048, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -13.22, 95% CI 2-sided [-26.32 to -0.13] — Week 20, Pain score
Statistical Analysis 44: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.102, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -13.23, 95% CI 2-sided [-29.11 to 2.64] — Week 24, Pain score
Statistical Analysis 45: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.030, MMRM — [p-value comment as in outcome 14, analysis 1]; Mean Difference (Net) = -16.70, 95% CI 2-sided [-31.79 to -1.62] — Week 24, Pain score

15. Secondary Outcome: Change From Baseline in Physical and Mental Component Scores (PCS, MCS) and in Domain Scores of Short Form 36 (SF-36) at All Assessment Time Points
Description: SF-36 is a generic health survey containing 36 questions covering 8 domains of health. SF-36 yields an 8-scale profile of functional health and well-being scores as well as PCS and MCS health summary scores. The version 2, 1-week recall questionnaire was used. Recoding, calculations and standardization were done as per the User's manual of SF-36. Domain scores were only calculated if less than half of the item scores were missing. All raw domain scores were transformed on a 0-100 scale (transformed domain scores) and then standardized into norm-based scores using Z-score. Following the transformation of the 8 domain scores into z-scores, the MCS and PCS were aggregated (AGG) using weights as PCS/MCS = 50 + (AGG_PHYS *10/AGG_MENT *10). High score (worse outcome) and low score (better outcome). Baseline was defined as the last available assessment prior to the start of study treatment. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline and Weeks 4, 12, 24
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | GSK3196165 22.5 mg | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 135 mg | GSK3196165 180 mg
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37 | 37
Scores on a scale
  PCS, Week 4,n=34,34,36,37,36,36,: number analyzed (Participants) | 34 | 34 | 36 | 37 | 36 | 36
  PCS, Week 4,n=34,34,36,37,36,36, | 1.86 (1.046) | 2.46 (1.048) | 5.05 (1.020) | 4.47 (1.007) | 4.80 (1.021) | 5.97 (1.028)
  PCS Week 12,n=34,35,35,37,35,36: number analyzed (Participants) | 34 | 35 | 35 | 37 | 35 | 36
  PCS Week 12,n=34,35,35,37,35,36 | 3.42 (1.203) | 4.88 (1.192) | 5.84 (1.186) | 5.15 (1.158) | 5.31 (1.188) | 6.97 (1.182)
  PCS, Week 24,n=8,14,21,24,19,34: number analyzed (Participants) | 8 | 14 | 21 | 24 | 19 | 34
  PCS, Week 24,n=8,14,21,24,19,34 | 5.34 (2.058) | 7.03 (1.631) | 6.63 (1.404) | 7.80 (1.335) | 7.50 (1.454) | 6.99 (1.211)
  MCS, Week 4,n=34,34,36,37,36,36,: number analyzed (Participants) | 34 | 34 | 36 | 37 | 36 | 36
  MCS, Week 4,n=34,34,36,37,36,36, | 3.36 (1.488) | 2.86 (1.488) | 3.81 (1.453) | 2.82 (1.434) | 4.52 (1.453) | 3.46 (1.453)
  MCS, Week 12,n=34,35,35,37,35,36,: number analyzed (Participants) | 34 | 35 | 35 | 37 | 35 | 36
  MCS, Week 12,n=34,35,35,37,35,36, | 3.54 (1.558) | 4.86 (1.542) | 5.00 (1.535) | 4.66 (1.501) | 5.51 (1.535) | 6.79 (1.521)
  MCS, Week 24,n=8,14,21,24,19,34: number analyzed (Participants) | 8 | 14 | 21 | 24 | 19 | 34
  MCS, Week 24,n=8,14,21,24,19,34 | 4.07 (2.560) | 4.50 (2.039) | 6.36 (1.755) | 3.02 (1.669) | 5.42 (1.817) | 7.86 (1.503)
  Bodily pain, Week 4,n=34,34,36,37,36,36,: number analyzed (Participants) | 34 | 34 | 36 | 37 | 36 | 36
  Bodily pain, Week 4,n=34,34,36,37,36,36, | 2.52 (1.071) | 2.41 (1.071) | 6.24 (1.043) | 5.44 (1.029) | 5.97 (1.046) | 7.60 (1.045)
  Bodily pain, Week 12,n=34,35,35,37,35,36: number analyzed (Participants) | 34 | 35 | 35 | 37 | 35 | 36
  Bodily pain, Week 12,n=34,35,35,37,35,36 | 3.90 (1.294) | 5.43 (1.280) | 6.72 (1.273) | 5.99 (1.243) | 6.01 (1.277) | 7.34 (1.263)
  Bodily pain, Week 24,n=8,14,21,24,19,34: number analyzed (Participants) | 8 | 14 | 21 | 24 | 19 | 34
  Bodily pain, Week 24,n=8,14,21,24,19,34 | 4.15 (2.580) | 7.01 (1.996) | 9.20 (1.682) | 7.36 (1.593) | 8.87 (1.752) | 9.35 (1.387)
  General Health, Week 4,n=34,34,36,37,36,36: number analyzed (Participants) | 34 | 34 | 36 | 37 | 36 | 36
  General Health, Week 4,n=34,34,36,37,36,36 | 1.78 (1.079) | 1.27 (1.079) | 2.77 (1.055) | 1.90 (1.039) | 3.43 (1.053) | 3.72 (1.054)
  General health, Week 12,n=34,35,35,37,35,36: number analyzed (Participants) | 34 | 35 | 35 | 37 | 35 | 36
  General health, Week 12,n=34,35,35,37,35,36 | 2.44 (1.102) | 3.07 (1.090) | 4.30 (1.088) | 3.02 (1.061) | 3.14 (1.087) | 4.73 (1.077)
  General health, Week 24,n=8,14,21,24,19,34: number analyzed (Participants) | 8 | 14 | 21 | 24 | 19 | 34
  General health, Week 24,n=8,14,21,24,19,34 | 2.07 (2.248) | 5.36 (1.762) | 4.83 (1.514) | 4.60 (1.420) | 3.84 (1.562) | 5.42 (1.265)
  Mental health, Week 4,n=34,34,36,37,36,36: number analyzed (Participants) | 34 | 34 | 36 | 37 | 36 | 36
  Mental health, Week 4,n=34,34,36,37,36,36 | 3.64 (1.451) | 3.77 (1.449) | 4.52 (1.413) | 3.62 (1.395) | 3.49 (1.413) | 3.69 (1.413)
  Mental health, Week 12,n=34,35,35,37,35,36: number analyzed (Participants) | 34 | 35 | 35 | 37 | 35 | 36
  Mental health, Week 12,n=34,35,35,37,35,36 | 2.27 (1.601) | 4.87 (1.581) | 5.49 (1.575) | 4.77 (1.539) | 4.68 (1.576) | 5.72 (1.558)
  Mental health, Week 24,n=8,14,21,24,19,34: number analyzed (Participants) | 8 | 14 | 21 | 24 | 19 | 34
  Mental health, Week 24,n=8,14,21,24,19,34 | 2.81 (2.619) | 4.13 (2.073) | 6.09 (1.777) | 3.42 (1.684) | 4.96 (1.844) | 7.82 (1.504)
  Physical functioning, Week 4,n=34,34,36,37,36,36: number analyzed (Participants) | 34 | 34 | 36 | 37 | 36 | 36
  Physical functioning, Week 4,n=34,34,36,37,36,36 | 3.30 (1.206) | 3.97 (1.208) | 5.68 (1.174) | 4.84 (1.159) | 5.18 (1.179) | 5.75 (1.180)
  Physical functioning, Week 12,n=34,35,35,37,35,36: number analyzed (Participants) | 34 | 35 | 35 | 37 | 35 | 36
  Physical functioning, Week 12,n=34,35,35,37,35,36 | 2.98 (1.390) | 5.80 (1.375) | 5.99 (1.368) | 5.98 (1.333) | 5.84 (1.373) | 7.76 (1.358)
  Physical functioning, Week 24,n=8,14,21,24,19,34: number analyzed (Participants) | 8 | 14 | 21 | 24 | 19 | 34
  Physical functioning, Week 24,n=8,14,21,24,19,34 | 6.93 (2.100) | 6.29 (1.700) | 6.52 (1.490) | 7.16 (1.426) | 7.40 (1.539) | 7.58 (1.309)
  Role emotional, Week 4,n=34,34,36,37,36,36: number analyzed (Participants) | 34 | 34 | 36 | 37 | 36 | 36
  Role emotional, Week 4,n=34,34,36,37,36,36 | 4.37 (1.489) | 3.09 (1.488) | 3.08 (1.452) | 3.35 (1.432) | 4.96 (1.451) | 3.77 (1.451)
  Role emotional, Week 12,n=34,35,35,37,35,36: number analyzed (Participants) | 34 | 35 | 35 | 37 | 35 | 36
  Role emotional, Week 12,n=34,35,35,37,35,36 | 4.85 (1.595) | 5.19 (1.574) | 5.52 (1.570) | 5.10 (1.532) | 5.93 (1.570) | 7.54 (1.552)
  Role emotional, Week 24,n=8,14,21,24,19,34: number analyzed (Participants) | 8 | 14 | 21 | 24 | 19 | 34
  Role emotional, Week 24,n=8,14,21,24,19,34 | 5.66 (2.674) | 6.57 (2.102) | 6.16 (1.794) | 4.36 (1.704) | 6.06 (1.863) | 8.18 (1.518)
  Role physical, Week 4,n=34,34,36,37,36,36: number analyzed (Participants) | 34 | 34 | 36 | 37 | 36 | 36
  Role physical, Week 4,n=34,34,36,37,36,36 | 2.15 (1.128) | 3.01 (1.124) | 4.04 (1.097) | 4.56 (1.082) | 4.02 (1.097) | 4.80 (1.099)
  Role physical, Week 12,n=34,35,35,37,35,36: number analyzed (Participants) | 34 | 35 | 35 | 37 | 35 | 36
  Role physical, Week 12,n=34,35,35,37,35,36 | 4.56 (1.270) | 5.16 (1.255) | 6.28 (1.251) | 5.49 (1.221) | 5.99 (1.253) | 7.91 (1.241)
  Role physical, Week 24,n=8,14,21,24,19,34: number analyzed (Participants) | 8 | 14 | 21 | 24 | 19 | 34
  Role physical, Week 24,n=8,14,21,24,19,34 | 6.38 (2.235) | 7.65 (1.738) | 6.27 (1.481) | 7.50 (1.408) | 7.59 (1.538) | 7.25 (1.250)
  Social functioning, Week 4,n=34,34,36,37,36,36: number analyzed (Participants) | 34 | 34 | 36 | 37 | 36 | 36
  Social functioning, Week 4,n=34,34,36,37,36,36 | 2.27 (1.512) | 1.95 (1.512) | 5.44 (1.475) | 2.84 (1.455) | 5.22 (1.476) | 5.67 (1.475)
  Social functioning, Week 12,n=34,35,35,37,35,36: number analyzed (Participants) | 34 | 35 | 35 | 37 | 35 | 36
  Social functioning, Week 12,n=34,35,35,37,35,36 | 4.34 (1.529) | 4.90 (1.513) | 4.34 (1.507) | 4.62 (1.471) | 6.32 (1.508) | 8.69 (1.491)
  Social functioning, Week 24,n=8,14,21,24,19,34: number analyzed (Participants) | 8 | 14 | 21 | 24 | 19 | 34
  Social functioning, Week 24,n=8,14,21,24,19,34 | 8.31 (2.841) | 5.41 (2.221) | 7.87 (1.871) | 4.52 (1.773) | 7.97 (1.951) | 8.60 (1.551)
  Vitality, Week 4,n=34,34,36,37,36,36: number analyzed (Participants) | 34 | 34 | 36 | 37 | 36 | 36
  Vitality, Week 4,n=34,34,36,37,36,36 | 1.91 (1.389) | 2.94 (1.386) | 5.48 (1.352) | 4.54 (1.334) | 6.55 (1.352) | 5.25 (1.353)
  Vitality, Week 12,n=34,35,35,37,35,36: number analyzed (Participants) | 34 | 35 | 35 | 37 | 35 | 36
  Vitality, Week 12,n=34,35,35,37,35,36 | 4.19 (1.445) | 6.16 (1.429) | 7.10 (1.421) | 6.37 (1.389) | 6.83 (1.421) | 8.16 (1.408)
  Vitality, Week 24,n=8,14,21,24,19,34: number analyzed (Participants) | 8 | 14 | 21 | 24 | 19 | 34
  Vitality, Week 24,n=8,14,21,24,19,34 | 4.68 (2.775) | 6.62 (2.175) | 7.83 (1.854) | 7.65 (1.758) | 8.04 (1.924) | 7.81 (1.560)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.683, MMRM — MMRM analysis adjusted for Baseline score, treatment group, visit and treatment group by visit and Baseline by visit interactions; Mean Difference (Net) = 0.60, 95% CI 2-sided [-2.31 to 3.52] — Week 4, PCS
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.030, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 3.19, 95% CI 2-sided [0.31 to 6.07] — Week 4, PCS
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.074, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 2.61, 95% CI 2-sided [-0.25 to 5.47] — Week 4, PCS
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.390, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 1.46, 95% CI 2-sided [-1.88 to 4.80] — Week 12, PCS
Statistical Analysis 5: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.154, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 2.42, 95% CI 2-sided [-0.91 to 5.75] — Week 12, PCS
Statistical Analysis 6: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.302, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 1.73, 95% CI 2-sided [-1.56 to 5.02] — Week 12, PCS
Statistical Analysis 7: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.521, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 1.69, 95% CI 2-sided [-3.50 to 6.88] — Week 24, PCS
Statistical Analysis 8: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.606, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 1.28, 95% CI 2-sided [-3.63 to 6.20] — Week 24, PCS
Statistical Analysis 9: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.320, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 2.46, 95% CI 2-sided [-2.41 to 7.32] — Week 24, PCS
Statistical Analysis 10: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.811, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = -0.50, 95% CI 2-sided [-4.65 to 3.64] — Week 4, MCS
Statistical Analysis 11: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.830, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 0.45, 95% CI 2-sided [-3.65 to 4.55] — Week 4, MCS
Statistical Analysis 12: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.795, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = -0.54, 95% CI 2-sided [-4.61 to 3.54] — Week 4, MCS
Statistical Analysis 13: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.548, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 1.32, 95% CI 2-sided [-3.00 to 5.64] — Week 12, MCS
Statistical Analysis 14: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.505, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 1.46, 95% CI 2-sided [-2.85 to 5.77] — Week 12, MCS
Statistical Analysis 15: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.605, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 1.12, 95% CI 2-sided [-3.15 to 5.39] — Week 12, MCS
Statistical Analysis 16: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.895, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 0.43, 95% CI 2-sided [-6.03 to 6.90] — Week 24, MCS
Statistical Analysis 17: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.461, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 2.29, 95% CI 2-sided [-3.84 to 8.42] — Week 24, MCS
Statistical Analysis 18: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.732, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = -1.05, 95% CI 2-sided [-7.10 to 4.99] — Week 24, MCS
Statistical Analysis 19: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.941, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = -0.11, 95% CI 2-sided [-3.11 to 2.88] — Week 4, Bodily Pain
Statistical Analysis 20: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.013, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 3.73, 95% CI 2-sided [0.78 to 6.67] — Week 4, Bodily Pain
Statistical Analysis 21: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.051, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 2.92, 95% CI 2-sided [-0.01 to 5.84] — Week 4, Bodily Pain
Statistical Analysis 22: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.403, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 1.53, 95% CI 2-sided [-2.07 to 5.12] — Week 12, Bodily Pain
Statistical Analysis 23: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.122, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 2.82, 95% CI 2-sided [-0.76 to 6.40] — Week 12, Bodily Pain
Statistical Analysis 24: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.247, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 2.08, 95% CI 2-sided [-1.45 to 5.62] — Week 12, Bodily Pain
Statistical Analysis 25: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.384, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 2.85, 95% CI 2-sided [-3.61 to 9.32] — Week 24, Bodily Pain
Statistical Analysis 26: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.105, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 5.05, 95% CI 2-sided [-1.07 to 11.16] — Week 24, Bodily Pain
Statistical Analysis 27: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.290, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 3.21, 95% CI 2-sided [-2.76 to 9.17] — Week 24, Bodily Pain
Statistical Analysis 28: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.738, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = -0.51, 95% CI 2-sided [-3.52 to 2.50] — Week 4, General Health
Statistical Analysis 29: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.513, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 0.99, 95% CI 2-sided [-1.99 to 3.97] — Week 4, General Health
Statistical Analysis 30: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.934, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 0.12, 95% CI 2-sided [-2.83 to 3.08] — Week 4, General Health
Statistical Analysis 31: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.687, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 0.63, 95% CI 2-sided [-2.43 to 3.68] — Week 12, General Health
Statistical Analysis 32: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.233, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 1.85, 95% CI 2-sided [-1.20 to 4.91] — Week 12, General Health
Statistical Analysis 33: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.708, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 0.57, 95% CI 2-sided [-2.44 to 3.59] — Week 12, General Health
Statistical Analysis 34: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.250, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 3.29, 95% CI 2-sided [-2.34 to 8.93] — Week 24, General Health
Statistical Analysis 35: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.307, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 2.76, 95% CI 2-sided [-2.57 to 8.09] — Week 24, General Health
Statistical Analysis 36: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.345, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 2.53, 95% CI 2-sided [-2.74 to 7.79] — Week 24, General Health
Statistical Analysis 37: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.950, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 0.16, 95% CI 2-sided [-0.19 to 0.52] — Week 4, Mental Health
Statistical Analysis 38: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.664, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 0.88, 95% CI 2-sided [-3.11 to 4.87] — Week 4, Mental Health
Statistical Analysis 39: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.994, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = -0.01, 95% CI 2-sided [-3.99 to 3.96] — Week 4, Mental Health
Statistical Analysis 40: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.250, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 2.60, 95% CI 2-sided [-1.84 to 7.03] — Week 12, Mental Health
Statistical Analysis 41: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.154, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 3.21, 95% CI 2-sided [-1.22 to 7.64] — Week 12, Mental Health
Statistical Analysis 42: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.262, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 2.50, 95% CI 2-sided [-1.88 to 6.89] — Week 12, Mental Health
Statistical Analysis 43: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.693, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 1.32, 95% CI 2-sided [-5.28 to 7.93] — Week 24, Mental Health
Statistical Analysis 44: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.302, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 3.28, 95% CI 2-sided [-2.98 to 9.54] — Week 24, Mental Health
Statistical Analysis 45: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.844, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 0.61, 95% CI 2-sided [-5.54 to 6.77] — Week 24, Mental Health
Statistical Analysis 46: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.698, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 0.66, 95% CI 2-sided [-2.71 to 4.04] — Week 4, Physical Functioning
Statistical Analysis 47: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.159, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 2.38, 95% CI 2-sided [-0.94 to 5.70] — Week 4, Physical Functioning
Statistical Analysis 48: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.360, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 1.53, 95% CI 2-sided [-1.76 to 4.83] — Week 4, Physical Functioning
Statistical Analysis 49: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.151, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 2.82, 95% CI 2-sided [-1.04 to 6.69] — Week 12, Physical Functioning
Statistical Analysis 50: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.124, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 3.01, 95% CI 2-sided [-0.83 to 6.86] — Week 12, Physical Functioning
Statistical Analysis 51: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.120, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 3.00, 95% CI 2-sided [-0.79 to 6.80] — Week 12, Physical Functioning
Statistical Analysis 52: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.814, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = -0.64, 95% CI 2-sided [-5.98 to 4.70] — Week 24, Physical Functioning
Statistical Analysis 53: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.873, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = -0.41, 95% CI 2-sided [-5.49 to 4.67] — Week 24, Physical Functioning
Statistical Analysis 54: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.928, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 0.23, 95% CI 2-sided [-4.80 to 5.26] — Week 24, Physical Functioning
Statistical Analysis 55: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.541, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = -1.29, 95% CI 2-sided [-5.44 to 2.86] — Week 4, Role Emotional
Statistical Analysis 56: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.535, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = -1.29, 95% CI 2-sided [-5.39 to 2.81] — Week 4, Role Emotional
Statistical Analysis 57: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.620, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = -1.03, 95% CI 2-sided [-5.10 to 3.05] — Week 4, Role Emotional
Statistical Analysis 58: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.881, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 0.34, 95% CI 2-sided [-4.08 to 4.76] — Week 12, Role Emotional
Statistical Analysis 59: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.767, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 0.66, 95% CI 2-sided [-3.74 to 5.07] — Week 12,Role Emotional
Statistical Analysis 60: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.913, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 0.24, 95% CI 2-sided [-4.12 to 4.61] — Week 12, Role Emotional
Statistical Analysis 61: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.790, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 0.91, 95% CI 2-sided [-5.81 to 7.63] — Week 24, Role Emotional
Statistical Analysis 62: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.876, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 0.50, 95% CI 2-sided [-5.86 to 6.87] — Week 24, Role Emotional
Statistical Analysis 63: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.684, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = -1.30, 95% CI 2-sided [-7.59 to 4.99] — Week 24, Role Emotional
Statistical Analysis 64: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.588, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 0.86, 95% CI 2-sided [-2.28 to 4.01] — Week 4, Role Physical
Statistical Analysis 65: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.229, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 1.90, 95% CI 2-sided [-1.21 to 5.00] — Week 4, Role Physical
Statistical Analysis 66: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.125, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 2.41, 95% CI 2-sided [-0.67 to 5.49] — Week 4, Role Physical
Statistical Analysis 67: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.736, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 0.60, 95% CI 2-sided [-2.92 to 4.12] — Week 12, Role Physical
Statistical Analysis 68: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.338, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 1.72, 95% CI 2-sided [-1.80 to 5.23] — Week 12, Role Physical
Statistical Analysis 69: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.600, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 0.92, 95% CI 2-sided [-2.55 to 4.40] — Week 12, Role Physical
Statistical Analysis 70: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.657, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 1.26, 95% CI 2-sided [-4.34 to 6.86] — Week 24, Role Physical
Statistical Analysis 71: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.965, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = -0.12, 95% CI 2-sided [-5.41 to 5.17] — Week 24, Role Physical
Statistical Analysis 72: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.675, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 1.12, 95% CI 2-sided [-4.14 to 6.37] — Week 24, Role Physical
Statistical Analysis 73: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.880, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = -0.32, 95% CI 2-sided [-4.54 to 3.89] — Week 4, Social Functioning
Statistical Analysis 74: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.135, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 3.17, 95% CI 2-sided [-1.00 to 7.33] — Week 4, Social Functioning
Statistical Analysis 75: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.785, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 0.57, 95% CI 2-sided [-3.56 to 4.71] — Week 4, Social Functioning
Statistical Analysis 76: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.797, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 0.55, 95% CI 2-sided [-3.69 to 4.80] — Week 12, Social Functioning
Statistical Analysis 77: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p > 0.999, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = -0.00, 95% CI 2-sided [-4.23 to 4.23] — Week 12, Social Functioning
Statistical Analysis 78: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.896, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 0.28, 95% CI 2-sided [-3.91 to 4.46] — Week 12, Social Functioning
Statistical Analysis 79: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.424, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = -2.89, 95% CI 2-sided [-10.02 to 4.24] — Week 24, Social Functioning
Statistical Analysis 80: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.898, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = -0.44, 95% CI 2-sided [-7.16 to 6.29] — Week 24, Social Functioning
Statistical Analysis 81: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.260, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = -3.79, 95% CI 2-sided [-10.42 to 2.84] — Week 24, Social Functioning
Statistical Analysis 82: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.603, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 1.02, 95% CI 2-sided [-2.85 to 4.90] — Week 4, Vitality
Statistical Analysis 83: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.068, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 3.56, 95% CI 2-sided [-0.26 to 7.39] — Week 4, Vitality
Statistical Analysis 84: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.174, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 2.63, 95% CI 2-sided [-1.17 to 6.43] — Week 4, Vitality
Statistical Analysis 85: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.334, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 1.97, 95% CI 2-sided [-2.04 to 5.98] — Week 12, Vitality
Statistical Analysis 86: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.153, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 2.91, 95% CI 2-sided [-1.09 to 6.91] — Week 12, Vitality
Statistical Analysis 87: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.279, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 2.18, 95% CI 2-sided [-1.78 to 6.13] — Week 12, Vitality
Statistical Analysis 88: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.584, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 1.94, 95% CI 2-sided [-5.04 to 8.91] — Week 24,Vitality
Statistical Analysis 89: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.346, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 3.15, 95% CI 2-sided [-3.44 to 9.73] — Week 24, Vitality
Statistical Analysis 90: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.370, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 2.97, 95% CI 2-sided [-3.55 to 9.48] — Week 24, Vitality
Statistical Analysis 91: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.045, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 2.94, 95% CI 2-sided [0.06 to 5.83] — Week 4, PCS
Statistical Analysis 92: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.006, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 4.11, 95% CI 2-sided [1.22 to 7.01] — Week 4, PCS
Statistical Analysis 93: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.264, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 1.89, 95% CI 2-sided [-1.44 to 5.23] — Week 12,PCS
Statistical Analysis 94: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.037, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 3.55, 95% CI 2-sided [0.22 to 6.88] — Week 12,PCS
Statistical Analysis 95: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.392, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 2.16, 95% CI 2-sided [-2.81 to 7.14] — Week 24, PCS
Statistical Analysis 96: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.493, MMRM — MMRM analysis adjusted for PCS Baseline score, treatment group, visit and treatment group by visit and Baseline by visit interactions; Mean Difference (Net) = 1.65, 95% CI 2-sided [-3.09 to 6.39] — Week 24, PCS
Statistical Analysis 97: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.577, MMRM — MMRM analysis adjusted for MCS Baseline score, treatment group, visit and treatment group by visit and Baseline by visit interactions; Mean Difference (Net) = 1.16, 95% CI 2-sided [-2.94 to 5.26] — Week 4, MCS
Statistical Analysis 98: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.964, MMRM — [p-value comment as in outcome 15, analysis 97]; Mean Difference (Net) = 0.10, 95% CI 2-sided [-4.01 to 4.20] — Week 4, MCS
Statistical Analysis 99: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.370, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 1.97, 95% CI 2-sided [-2.35 to 6.28] — Week 12, MCS
Statistical Analysis 100: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.138, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 3.25, 95% CI 2-sided [-1.05 to 7.54] — Week 12, MCS
Statistical Analysis 101: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.667, MMRM — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Net) = 1.36, 95% CI 2-sided [-4.85 to 7.56] — Week 24, MCS
Statistical Analysis 102: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.203, MMRM — MMRM analysis adjusted for Baseline, treatment group, visit, treatment group by visit and Baseline by visit interactions; Mean Difference (Net) = 3.79, 95% CI 2-sided [-4.85 to 7.56] — Week 24, MCS
Statistical Analysis 103: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.023, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 3.45, 95% CI 2-sided [0.49 to 6.41] — Week 4, Bodily pain
Statistical Analysis 104: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p < 0.001, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 5.08, 95% CI 2-sided [2.14 to 8.03] — Week 4, Bodily pain
Statistical Analysis 105: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.249, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 2.11, 95% CI 2-sided [-1.49 to 5.70] — Week 12, Bodily pain
Statistical Analysis 106: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.059, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 3.43, 95% CI 2-sided [-0.13 to 6.99] — Week 12, Bodily pain
Statistical Analysis 107: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.134, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 4.72, 95% CI 2-sided [-1.47 to 10.90] — Week 24, Bodily pain
Statistical Analysis 108: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.078, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 5.20, 95% CI 2-sided [-0.58 to 10.97] — Week 24, Bodily pain
Statistical Analysis 109: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.275, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 1.65, 95% CI 2-sided [-1.32 to 4.62] — Week 4, General health
Statistical Analysis 110: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.199, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 1.94, 95% CI 2-sided [-1.03 to 4.91] — Week 4, General health
Statistical Analysis 111: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.654, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 0.69, 95% CI 2-sided [-2.36 to 3.74] — Week 12, General health
Statistical Analysis 112: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.138, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 2.29, 95% CI 2-sided [-0.74 to 5.33] — Week 12, General health
Statistical Analysis 113: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.516, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 1.77, 95% CI 2-sided [-3.62 to 7.17] — Week 24, General health
Statistical Analysis 114: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.198, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 3.35, 95% CI 2-sided [-1.77 to 8.46] — Week 24, General health
Statistical Analysis 115: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.941, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = -0.15, 95% CI 2-sided [-4.15 to 3.84] — Week 4, Mental health
Statistical Analysis 116: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.979, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 0.05, 95% CI 2-sided [-3.94 to 4.05] — Week 4, Mental health
Statistical Analysis 117: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.287, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 2.40, 95% CI 2-sided [-2.03 to 6.84] — Week 12, Mental health
Statistical Analysis 118: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.125, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 3.45, 95% CI 2-sided [-0.96 to 7.85] — Week 12, Mental health
Statistical Analysis 119: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.503, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 2.15, 95% CI 2-sided [-4.18 to 8.49] — Week 24, Mental health
Statistical Analysis 120: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.099, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 5.01, 95% CI 2-sided [-0.96 to 10.98] — Week 24,Mental health
Statistical Analysis 121: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.268, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 1.88, 95% CI 2-sided [-1.45 to 5.21] — Week 4, Physical functioning
Statistical Analysis 122: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.147, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 2.45, 95% CI 2-sided [-0.87 to 5.77] — Week 4, Physical functioning
Statistical Analysis 123: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.145, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 2.87, 95% CI 2-sided [-0.99 to 6.73] — Week 12, Physical functioning
Statistical Analysis 124: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.014, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 2.54, 95% CI 2-sided [0.97 to 8.61] — Week 12, Physical functioning
Statistical Analysis 125: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.856, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 0.47, 95% CI 2-sided [-4.66 to 5.61] — Week 24, Physical functioning
Statistical Analysis 126: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.793, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 0.65, 95% CI 2-sided [-4.24 to 5.55] — Week 24, Physical functioning
Statistical Analysis 127: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.778, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 0.59, 95% CI 2-sided [-3.51 to 4.69] — Week 4, Role emotional
Statistical Analysis 128: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.773, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = -0.60, 95% CI 2-sided [-4.70 to 3.50] — Week 4, Role emotional
Statistical Analysis 129: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.631, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 1.08, 95% CI 2-sided [-3.34 to 5.49] — Week 12, Role emotional
Statistical Analysis 130: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.230, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 2.68, 95% CI 2-sided [-1.71 to 7.07] — Week 12, Role emotional
Statistical Analysis 131: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.901, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 0.41, 95% CI 2-sided [-6.03 to 6.84] — Week 24, Role emotional
Statistical Analysis 132: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.412, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 2.52, 95% CI 2-sided [-3.54 to 8.59] — Week 24, Role emotional
Statistical Analysis 133: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.234, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 1.88, 95% CI 2-sided [-1.22 to 4.98] — Week 4, Role physical
Statistical Analysis 134: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.094, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 2.66, 95% CI 2-sided [-0.46 to 5.77] — Week 4, Role physical
Statistical Analysis 135: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.423, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 1.43, 95% CI 2-sided [-2.08 to 4.94] — Week 12, Role physical
Statistical Analysis 136: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.061, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 3.35, 95% CI 2-sided [-0.16 to 6.86] — Week 12, Role physical
Statistical Analysis 137: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.657, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 1.21, 95% CI 2-sided [-4.16 to 6.57] — Week 24, Role physical
Statistical Analysis 138: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.737, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 0.87, 95% CI 2-sided [-4.22 to 5.95] — Week 24, Role physical
Statistical Analysis 139: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.165, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 2.95, 95% CI 2-sided [-1.22 to 7.11] — Week 4, Social Functioning
Statistical Analysis 140: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.109, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 3.40, 95% CI 2-sided [-0.77 to 7.56] — Week 4, Social Functioning
Statistical Analysis 141: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.359, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 1.98, 95% CI 2-sided [-2.26 to 6.21] — Week 12, Social Functioning
Statistical Analysis 142: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.043, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 4.35, 95% CI 2-sided [0.14 to 8.56] — Week 12, Social Functioning
Statistical Analysis 143: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.923, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = -0.33, 95% CI 2-sided [-7.15 to 6.49] — Week 24, Social Functioning
Statistical Analysis 144: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.927, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 0.30, 95% CI 2-sided [-6.11 to 6.70] — Week 24, Social Functioning
Statistical Analysis 145: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.018, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 4.64, 95% CI 2-sided [0.82 to 8.46] — Week 4, Vitality
Statistical Analysis 146: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.087, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 3.34, 95% CI 2-sided [-0.49 to 7.17] — Week 4, Vitality
Statistical Analysis 147: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.193, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 2.64, 95% CI 2-sided [-1.35 to 6.64] — Week 12, Vitality
Statistical Analysis 148: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.051, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 3.97, 95% CI 2-sided [-0.01 to 7.95] — Week 12, Vitality
Statistical Analysis 149: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.321, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 3.36, 95% CI 2-sided [-3.31 to 10.02] — Week 24, Vitality
Statistical Analysis 150: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.328, MMRM — [p-value comment as in outcome 15, analysis 102]; Mean Difference (Net) = 3.13, 95% CI 2-sided [-3.18 to 9.44] — Week 24, Vitality

16. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue at All Assessment Time Points
Description: The FACIT-fatigue questionnaire is a participant reported measure developed to assess fatigue consisting of 13 statements regarding feeling fatigue using a numeric rating scale ranging from 0 to 4. For only two of the items (i.e. Answer 5 [An5] and An7) a higher value represents a lower fatigue; 11 of the item scores (i.e. HI7, HI12, An1, An2, An3, An4, An8, An12, An14, An15, An16) have to be reversed by subtracting the captured value from 4 (0 is turned to a 4; 1 into 3; 3 into 1; 4 into 0). After performing the reversals the sum of the non-missing individual items were multiplied by 13 and divided by the number of the non-missing individual items. The final score ranges from 0 to 52 with higher values representing a lower fatigue (i.e. a better quality of life). Baseline was defined as the last available assessment prior to the start of study treatment. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline and Weeks 4, 12, 24
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | GSK3196165 22.5 mg | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 135 mg | GSK3196165 180 mg
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37 | 37
Scores on a scale
  Week 4,n=34,34,36,37, 36, 36: number analyzed (Participants) | 34 | 34 | 36 | 37 | 36 | 36
  Week 4,n=34,34,36,37, 36, 36 | 3.16 (1.192) | 2.51 (1.191) | 4.66 (1.164) | 5.71 (1.148) | 6.73 (1.165) | 5.97 (1.165)
  Week 12,n=34,35,35,37, 35, 36: number analyzed (Participants) | 34 | 35 | 35 | 37 | 35 | 36
  Week 12,n=34,35,35,37, 35, 36 | 3.37 (1.291) | 5.29 (1.278) | 5.91 (1.273) | 6.44 (1.244) | 7.28 (1.274) | 8.70 (1.262)
  Week 24,n=8,14,21,24, 19, 34: number analyzed (Participants) | 8 | 14 | 21 | 24 | 19 | 34
  Week 24,n=8,14,21,24, 19, 34 | 7.56 (2.439) | 8.31 (1.946) | 7.09 (1.680) | 6.74 (1.595) | 8.28 (1.737) | 9.43 (1.443)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.701, MMRM — MMRM analysis adjusted for FACIT Baseline score, treatment group, visit and treatment group by visit and Baseline by visit interactions; Mean Difference (Net) = -0.65, 95% CI 2-sided [-3.97 to 2.67] — Week 4, FACIT score
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.370, MMRM — [p-value comment as in outcome 16, analysis 1]; Mean Difference (Net) = 1.50, 95% CI 2-sided [-1.79 to 4.78] — Week 4, FACIT score
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.125, MMRM — [p-value comment as in outcome 16, analysis 1]; Mean Difference (Net) = 2.55, 95% CI 2-sided [-0.71 to 5.81] — Week 4, FACIT score
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.292, MMRM — [p-value comment as in outcome 16, analysis 1]; Mean Difference (Net) = 1.92, 95% CI 2-sided [-1.66 to 5.50] — Week 12, FACIT score
Statistical Analysis 5: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.163, MMRM — [p-value comment as in outcome 16, analysis 1]; Mean Difference (Net) = 6.11, 95% CI 2-sided [-1.04 to 6.11] — Week 12, FACIT sscore
Statistical Analysis 6: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.087, MMRM — [p-value comment as in outcome 16, analysis 1]; Mean Difference (Net) = 3.08, 95% CI 2-sided [-0.46 to 6.61] — Week 12, FACIT score
Statistical Analysis 7: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.808, MMRM — [p-value comment as in outcome 16, analysis 1]; Mean Difference (Net) = 0.76, 95% CI 2-sided [-5.40 to 6.92] — Week 24, FACIT score
Statistical Analysis 8: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.874, MMRM — [p-value comment as in outcome 16, analysis 1]; Mean Difference (Net) = -0.47, 95% CI 2-sided [-6.31 to 5.38] — Week 24, FACIT score
Statistical Analysis 9: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.780, MMRM — [p-value comment as in outcome 16, analysis 1]; Mean Difference (Net) = -0.81, 95% CI 2-sided [-6.58 to 4.95] — Week 24,FACIT score
Statistical Analysis 10: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.033, MMRM — [p-value comment as in outcome 16, analysis 1]; Mean Difference (Net) = 3.57, 95% CI 2-sided [0.29 to 6.85] — Week 4, FACIT score
Statistical Analysis 11: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.094, MMRM — [p-value comment as in outcome 16, analysis 1]; Mean Difference (Net) = 2.81, 95% CI 2-sided [-0.48 to 6.10] — Week 4, FACIT score
Statistical Analysis 12: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.032, MMRM — [p-value comment as in outcome 16, analysis 1]; Mean Difference (Net) = 3.92, 95% CI 2-sided [0.34 to 7.49] — Week 12, FACIT score
Statistical Analysis 13: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.004, MMRM — [p-value comment as in outcome 16, analysis 1]; Mean Difference (Net) = 5.33, 95% CI 2-sided [1.77 to 8.89] — Week 12, FACIT score
Statistical Analysis 14: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.808, MMRM — [p-value comment as in outcome 16, analysis 1]; Mean Difference (Net) = 0.73, 95% CI 2-sided [-5.19 to 6.64] — Week 24, FACIT score
Statistical Analysis 15: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.511, MMRM — [p-value comment as in outcome 16, analysis 1]; Mean Difference (Net) = 1.87, 95% CI 2-sided [-3.74 to 7.48] — Week 24, FACIT score

17. Secondary Outcome: Change From Baseline in Brief Fatigue Inventory (BFI) Question 3 at All Assessment Time Points
Description: BFI is a self-reported instrument consisting of nine questions which correlate well with quality-of-life measures. For this study, Question 3 only was used which asked about fatigue severity at its worst in the last 24 hours. A discrete 11 unit numeric reporting scale was used where 0 =No fatigue, and 10=As bad as you can imagine. Baseline was defined as the last available assessment prior to the start of study treatment. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline and Weeks 4, 12, 24
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | GSK3196165 22.5 mg | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 135 mg | GSK3196165 180 mg
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37 | 37
Scores on a scale
  Week 4,n=34,34,36,37, 36, 36: number analyzed (Participants) | 34 | 34 | 36 | 37 | 36 | 36
  Week 4,n=34,34,36,37, 36, 36 | -0.60 (0.348) | -0.67 (0.348) | -1.10 (0.339) | -1.60 (0.335) | -1.86 (0.339) | -1.53 (0.341)
  Week 12,n=34,35,35,37, 35, 36: number analyzed (Participants) | 34 | 35 | 35 | 37 | 35 | 36
  Week 12,n=34,35,35,37, 35, 36 | -0.63 (0.346) | -1.26 (0.342) | -1.83 (0.341) | -2.02 (0.333) | -2.07 (0.341) | -2.20 (0.339)
  Week 24,n=8,14,21,24, 19, 34: number analyzed (Participants) | 8 | 14 | 21 | 24 | 19 | 34
  Week 24,n=8,14,21,24, 19, 34 | -1.83 (0.635) | -2.19 (0.496) | -1.76 (0.418) | -2.03 (0.395) | -2.59 (0.435) | -2.41 (0.353)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.888, MMRM — MMRM analysis adjusted for BFI Baseline score, treatment group, visit and treatment group by visit and Baseline by visit interactions; Mean Difference (Net) = -0.07, 95% CI 2-sided [-1.04 to 0.90] — Week 4, BFI score
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.307, MMRM — [p-value comment as in outcome 17, analysis 1]; Mean Difference (Net) = -0.50, 95% CI 2-sided [-1.46 to 0.46] — Week 4, BFI score
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.041, MMRM — [p-value comment as in outcome 17, analysis 1]; Mean Difference (Net) = -0.99, 95% CI 2-sided [-1.95 to -0.04] — Week 4, BFI score
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.191, MMRM — [p-value comment as in outcome 17, analysis 1]; Mean Difference (Net) = -0.64, 95% CI 2-sided [-1.60 to 0.32] — Week 12, BFI score
Statistical Analysis 5: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.014, MMRM — [p-value comment as in outcome 17, analysis 1]; Mean Difference (Net) = -1.20, 95% CI 2-sided [-2.16 to -0.24] — Week 12, BFI score
Statistical Analysis 6: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.004, MMRM — [p-value comment as in outcome 17, analysis 1]; Mean Difference (Net) = -1.39, 95% CI 2-sided [-2.34 to -0.45] — Week 12, BFI score
Statistical Analysis 7: Comparison: Placebo vs GSK3196165 22.5 mg; Test type: Other; p = 0.656, MMRM — [p-value comment as in outcome 17, analysis 1]; Mean Difference (Net) = -0.36, 95% CI 2-sided [-1.94 to 1.23] — Week 24, BFI score
Statistical Analysis 8: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; p = 0.928, MMRM — [p-value comment as in outcome 17, analysis 1]; Mean Difference (Net) = 0.07, 95% CI 2-sided [-1.43 to 1.57] — Week 24, BFI score
Statistical Analysis 9: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; p = 0.788, MMRM — [p-value comment as in outcome 17, analysis 1]; Mean Difference (Net) = -0.20, 95% CI 2-sided [-1.68 to 1.28] — Week 24, BFI score
Statistical Analysis 10: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.010, MMRM — [p-value comment as in outcome 17, analysis 1]; Mean Difference (Net) = -1.26, 95% CI 2-sided [-2.22 to -0.30] — Week 4, BFI score
Statistical Analysis 11: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.059, MMRM — [p-value comment as in outcome 17, analysis 1]; Mean Difference (Net) = -0.93, 95% CI 2-sided [-1.89 to 0.03] — Week 4, BFI score
Statistical Analysis 12: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.003, MMRM — [p-value comment as in outcome 17, analysis 1]; Mean Difference (Net) = -1.44, 95% CI 2-sided [-2.40 to -0.48] — Week 12, BFI score
Statistical Analysis 13: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.001, MMRM — [p-value comment as in outcome 17, analysis 1]; Mean Difference (Net) = -1.57, 95% CI 2-sided [-2.53 to -0.62] — Week 12, BFI score
Statistical Analysis 14: Comparison: Placebo vs GSK3196165 135 mg; Test type: Other; p = 0.324, MMRM — [p-value comment as in outcome 17, analysis 1]; Mean Difference (Net) = -0.76, 95% CI 2-sided [-2.28 to 0.76] — Week 24, BFI score
Statistical Analysis 15: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; p = 0.432, MMRM — [p-value comment as in outcome 17, analysis 1]; Mean Difference (Net) = -0.58, 95% CI 2-sided [-2.02 to 0.87] — Week 24, BFI score

18. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious AEs (SAEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participants, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, is associated with liver injury and impaired liver function or any other situations as per Medical or Scientific judgment. Overall AEs and SAEs for the entire study duration until follow-up have been presented.
Time Frame: Up to 62 weeks
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3196165 22.5 mg | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 135 mg | GSK3196165 180 mg
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37 | 37
Participants
  Any AE | 26 | 24 | 26 | 28 | 28 | 24
  Any SAE | 1 | 2 | 1 | 2 | 2 | 0

19. Secondary Outcome: Number of Participants With Serious Infections
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participants, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Serious infections were categorized as AE of special interest. The number of participants with overall serious infections have been presented.
Time Frame: Up to 62 weeks
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3196165 22.5 mg | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 135 mg | GSK3196165 180 mg
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37 | 37
Participants | 0 | 1 | 0 | 0 | 0 | 0

20. Secondary Outcome: Number of Participants With Opportunistic Infections
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participants, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Opportunistic infections were categorized as AE of special interest. The number of participants with overall opportunistic infections have been presented.
Time Frame: Up to 62 weeks
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3196165 22.5 mg | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 135 mg | GSK3196165 180 mg
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37 | 37
Participants | 0 | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Number of Participants With Pulmonary Events
Description: Pulmonary assessments were performed to determine the number of participants with pulmonary events including persistent cough, persistent dyspnea, and persistent Diffusing capacity of the lung for carbon monoxide (DLCO). Persistent is defined as any event with duration >=15 days. Baseline was defined as the last available assessment prior to the start of study treatment. The number of participants experiencing pulmonary events have been reported.
Time Frame: Up to 62 weeks
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3196165 22.5 mg | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 135 mg | GSK3196165 180 mg
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37 | 37
Participants
  Persistent Cough | 1 | 0 | 0 | 0 | 0 | 0
  Persistent Dyspnea | 1 | 0 | 0 | 1 | 0 | 0
  Persistent DLCO decrease >15% from Baseline | 2 | 3 | 1 | 0 | 3 | 1

22. Secondary Outcome: Number of Participants With Worst-case Post-Baseline Results for Pulse Oximetry
Description: Oxygen saturation measures the capacity of blood to transport oxygen to other parts of the body. Oxygen binds to hemoglobin in red blood cells when moving through the lungs. A pulse oximeter uses two frequencies of light (red and infrared) to determine the percentage of hemoglobin in the blood that is saturated with oxygen, that is called as blood oxygen saturation. Baseline was defined as the last available assessment prior to the start of study treatment. The number of participants with blood oxygen level < 80%, 80% to <90% and >=90% have been reported.
Time Frame: Up to 62 weeks
Population: ITT Population. Only those participants with data available at specified time point were analyzed (represented by n=x in category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3196165 22.5 mg | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 135 mg | GSK3196165 180 mg
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37 | 37
Participants
  < 80%; n=37, 36, 37, 37, 36, 37: number analyzed (Participants) | 37 | 36 | 37 | 37 | 36 | 37
  < 80%; n=37, 36, 37, 37, 36, 37 | 0 | 0 | 0 | 0 | 0 | 0
  80% to <90%; n=37, 36, 37, 37, 36, 37: number analyzed (Participants) | 37 | 36 | 37 | 37 | 36 | 37
  80% to <90%; n=37, 36, 37, 37, 36, 37 | 0 | 0 | 0 | 0 | 1 | 0
  >= 90%; n=37, 36, 37, 37, 36, 37: number analyzed (Participants) | 37 | 36 | 37 | 37 | 36 | 37
  >= 90%; n=37, 36, 37, 37, 36, 37 | 37 | 36 | 37 | 37 | 35 | 37

ADVERSE EVENTS:
Time Frame: Up to 62 weeks
Description: ITT Population was used for the analysis of safety data.
Groups:
- Placebo: Participants received placebo liquid (sterile 0.9% weight/volume) sodium chloride solution) 0.6 mL drawn into a small (1 mL syringe) administered subcutaneous in the thigh/abdomen up to 52 weeks in combination with MTX tablets (orally)/liquid (subcutaneous injection) at a dose of 7.5 to 25 mg/week and folic acid tablet/capsule (orally) at a dose of >=5 mg/week. MTX was taken as a single weekly dose/divided weekly dose, folic acid was taken the day after and at least 12 hours following MTX administration. Safety was monitored for 1 hour after the injection, for the first 3 injections, then for 30 minutes thereafter.
- GSK3196165 22.5 mg: Participants received GSK3196165 22.5 mg (0.15 mL) liquid drawn into a small (03 ml/0.5 ml syringe) administered subcutaneous in the thigh/abdomen up to 52 weeks in combination with MTX tablets (orally)/liquid (subcutaneous injection) at a dose of 7.5 to 25 mg/week and folic acid tablet/capsule (orally) at a dose of >=5 mg/week. MTX was taken as a single weekly dose/divided weekly dose, folic acid was taken the day after and at least 12 hours following MTX administration. Safety was monitored for 1 hour after the injection, for the first 3 injections, then for 30 minutes thereafter.
- GSK3196165 45 mg: Participants received GSK3196165 45 mg (0.3 mL) liquid drawn into a small (03 ml/0.5 ml syringe) administered subcutaneous in the thigh/abdomen up to 52 weeks in combination with MTX tablets (orally)/liquid (subcutaneous injection) at a dose of 7.5 to 25 mg/week and folic acid tablet/capsule (orally) at a dose of >=5 mg/week. MTX was taken as a single weekly dose/divided weekly dose, folic acid was taken the day after and at least 12 hours following MTX administration. Safety was monitored for 1 hour after the injection, for the first 3 injections, then for 30 minutes thereafter.
- GSK3196165 90 mg: Participants received GSK3196165 90 mg (0.6 mL) liquid drawn into a small (1 ml syringe) administered subcutaneous in the thigh/abdomen up to 52 weeks in combination with MTX tablets (orally)/liquid (subcutaneous injection) at a dose of 7.5 to 25 mg/week and folic acid tablet/capsule (orally) at a dose of >=5 mg/week. MTX was taken as a single weekly dose/divided weekly dose, folic acid was taken the day after and at least 12 hours following MTX administration. Safety was monitored for 1 hour after the injection, for the first 3 injections, then for 30 minutes thereafter.
- GSK3196165 135 mg: Participants received GSK3196165 135 mg (0.9 mL) liquid drawn into a small (1 ml syringe) administered subcutaneous in the thigh/abdomen up to 52 weeks in combination with MTX tablets (orally)/liquid (subcutaneous injection) at a dose of 7.5 to 25 mg/week and folic acid tablet/capsule (orally) at a dose of >=5 mg/week. MTX was taken as a single weekly dose/divided weekly dose, folic acid was taken the day after and at least 12 hours following MTX administration. Safety was monitored for 1 hour after the injection, for the first 3 injections, then for 30 minutes thereafter.
Arm/Group | Placebo | GSK3196165 22.5 mg | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 135 mg | GSK3196165 180 mg
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/37 | 0/37 | 0/37 | 0/37 | 0/37
Serious Adverse Events (participants affected / at risk) | 1/37 | 2/37 | 1/37 | 2/37 | 2/37 | 0/37
Other Adverse Events (participants affected / at risk) | 13/37 | 12/37 | 13/37 | 9/37 | 18/37 | 13/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=37) | GSK3196165 22.5 mg (N=37) | GSK3196165 45 mg (N=37) | GSK3196165 90 mg (N=37) | GSK3196165 135 mg (N=37) | GSK3196165 180 mg (N=37)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=37) | GSK3196165 22.5 mg (N=37) | GSK3196165 45 mg (N=37) | GSK3196165 90 mg (N=37) | GSK3196165 135 mg (N=37) | GSK3196165 180 mg (N=37)
Nasopharyngitis (Infections and infestations) | 8 (8) | 5 (6) | 7 (11) | 5 (6) | 8 (8) | 9 (12)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 5 (6) | 3 (3) | 2 (2) | 7 (9) | 3 (4)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 3 (5) | 5 (5)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 3 (8) | 3 (3) | 3 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-03-11): https://cdn.clinicaltrials.gov/large-docs/71/NCT02504671/Prot_000.pdf
  • Statistical Analysis Plan (2015-08-26): https://cdn.clinicaltrials.gov/large-docs/71/NCT02504671/SAP_001.pdf